## STATISTICAL ANALYSIS PLAN

A multi-center, randomized, double-blind, placebo-controlled, parallel group-comparison trial to assess the efficacy and safety of brexpiprazole as adjunctive therapy in patients with major depressive disorder

NCT Number: NCT03697603

PRT NO.: 331-102-00058

Version Date: 10 Aug 2022 (Version 1.0)

## Otsuka Pharmaceutical Co., Ltd.

Investigational New Drug Brexpiprazole (OPC-34712)

Protocol No. 331-102-00058

A multi-center, randomized, double-blind, placebo-controlled, parallel group-comparison trial to assess the efficacy and safety of brexpiprazole as adjunctive therapy in patients with major depressive disorder

Statistical Analysis Plan

Version: 1.0
Date: 10 Aug 2022
Protocol Version 3 Date: 23 Jan 2020

Confidential
May not be used, divulged, published, or otherwise disclosed without the prior written consent of Otsuka Pharmaceutical Co., Ltd.

## **Table of Contents**

| Tabl | Table of Contents | |
|---|---|---|
| List | of Appendices | 5 |
| List | of Abbreviations and Definition of Terms | 6 |
| 1 | Introduction | 8 |
| 2 | Trial Objectives | |
| 3 | Trial Design | |
| 3.1 | Type/Design of Trial | |
| 3.2 | Trial Treatments | 9 |
| 3.2.1 | Antidepressant Treatment Period (Phase A) | 9 |
| 3.2.2 | Double-blind Period (Phase B) | 10 |
| 3.2.3 | Antidepressant-responder Treatment-continuation Period (Phase A+) | 11 |
| 3.3 | Trial Population | 11 |
| 3.3.1 | Number of Subjects and Trial Population | 11 |
| 3.4 | Trial Visit Window | 12 |
| 3.5 | Handling of Endpoints | 13 |
| 3.5.1 | Montgomery Åsberg Depression Rating Scale (MADRS) | 13 |
| 3.5.2 | Clinical Global Impression – Improvement (CGI-I) | 13 |
| 3.5.3 | Clinical Global Impression - Severity of Illness (CGI-S) | 13 |
| 3.5.4 | Hamilton Rating Scale for Depression (HAM-D) | 13 |
| 3.5.5 | Sheehan Disability Scale (SDS) | 13 |
| 3.5.6 | Montgomery Åsberg Depression Rating Scale Self-assessment (MADRS-S) | 14 |
| 3.5.7 | Drug-induced Extrapyramidal Symptoms Scale (DIEPSS) | 14 |
| 3.5.8 | Abnormal Involuntary Movement Scale (AIMS) | 14 |
| 4 | Sample Size | 14 |
| 5 | Statistical Analysis Datasets | 14 |
| 5.1 | Pharmacokinetic Analysis Set | 14 |
| 5.2 | Full Analysis Set | 15 |
| 5.3 | Safety Analysis Set | 15 |
| 5.4 | Antidepressant Therapy Set | 15 |

| 5.5 | Phase A+ Set | 15 |
|---|---|---|
| 5.6 | Handling of Missing Data | |
| 6 | Primary and Secondary Outcome Variables: | 15 |
| 6.1 | Primary Outcome Variables | |
| 6.2 | Secondary Outcome Variables | 16 |
| 7 | Disposition and Demographic Analysis | 16 |
| 7.1 | Subject Disposition | |
| 7.2 | Demographic and Baseline Characteristics | 17 |
| 7.3 | Baseline Disease Evaluation | 17 |
| 7.4 | Treatment Compliance | 18 |
| 7.5 | Prior and Concomitant Medications | 18 |
| 7.6 | Protocol Deviations | 19 |
| 8 | Efficacy Analysis | 19 |
| 8.1 | Primary Efficacy Endpoint | 19 |
| 8.1.1 | Primary Efficacy Analysis | 19 |
| 8.1.2 | Sensitivity Analyses | 20 |
| 8.1.2.1 | Sensitivity Analysis for Handling of Missing Data | 20 |
| 8.1.2.2 | Sensitivity Analysis for Normality Assumption | 21 |
| 8.1.3 | Technical Computational Details for Primary Efficacy Analysis | 21 |
| 8.2 | Secondary Efficacy Analyses | 21 |
| 8.3 | Subgroup Analyses | 22 |
| 8.4 | Exploratory or Other Analyses | 23 |
| 9 | Safety Analyses | 23 |
| 9.1 | Extent of Exposure | 24 |
| 9.2 | Adverse Events | 24 |
| 9.2.1 | Adverse Events of Interest | 25 |
| 9.2.2 | Subgroup Analysis of Adverse Events | 25 |
| 9.2.3 | Adverse Events in the Antidepressant Treatment Period (Phase A) and the Antidepressant-responder Treatment-continuation Period (Phase A+) | 26 |
| 9.3 | Clinical Laboratory Data | |
| 9.4 | Vital Sign Data | |

## Protocol 331-102-00058

| 9.5 | Physical Examination Data | 29 |
|-------|--------------------------------------------------------|----|
| 9.6 | Electrocardiogram Data | 29 |
| 9.7 | Other Safety Data | 30 |
| 9.7.1 | Body Weight, BMI, and Waist Circumference | 30 |
| 9.7.2 | DIEPSS, AIMS, and Barnes Akathisia Rating Scale (BARS) | 30 |
| 9.7.3 | Columbia-Suicide Severity Rating Scale (C-SSRS) | 31 |
| 10 | Pharmacokinetic Analyses | 32 |
| 11 | Pharmacodynamic Analyses | 32 |
| 12 | Pharmacogenomic Analyses | 32 |
| 13 | Interim Analysis | 33 |
| 14 | Changes in the Planned Analyses | 33 |
| 15 | References | 33 |

## **List of Appendices**

| Appendix 1 | Criteria for Identifying Vital Signs and Weight of Potential Clinical Relevance | 34 |
|---|---|---|
| Appendix 2 | Criteria for Identifying Laboratory Values of Potential Clinical Relevance | 35 |
| Appendix 3 | Criteria for Identifying ECG Measurements of Potential Clinical Relevance | 36 |
| Appendix 4 | Adverse Events of Interest | 37 |
| Appendix 5 | List of Summary Tables | 94 |
| Appendix 6 | List of Subject Data Listings | 104 |

## **List of Abbreviations and Definition of Terms**

| <b>Abbreviation</b> | <u>Definition</u> |
|---|---|
| ADT | Antidepressant therapy |
| AIMS | Abnormal Involuntary Movement Scale |
| ALT | Alanine aminotransferase |
| ANCOVA | Analysis of covariance |
| AST | Aspartate aminotransferase |
| BARS | Barnes Akathisia Rating Scale Barnes |
| BMI | Body mass index |
| BUN | Blood urea nitrogen |
| CGI | Clinical Global Impression |
| CGI-I | Clinical Global Impression - Improvement |
| CGI-S | Clinical Global Impression - Severity of Illness |
| CMH | Cochran-Mantel-Haenszel |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CYP | Cytochrome P450 |
| DIEPSS | Drug Induced Extra-Pyramidal Symptoms Scale |
| DSM-5 | Diagnostic and statistical manual of mental disorders fifth edition |
| EM | Extensive metabolizer |
| GOT | Glutamic-oxaloacetic transaminase |
| GPT | Glutamic-pyruvic transaminase |
| FAS | Full analysis set |
| HAM-D | Hamilton Rating Scale for Depression |
| HDL | High-density lipoprotein |
| IM | Intermediate metabolizer |
| IMP | Investigational medicinal product |
| LDL | Low-density lipoprotein |
| LOCF | Last observation carried forward |
| MADRS | Montgomery Åsberg Depression Rating Scale |
| MADRS-S | The Montgomery Asberg Depression Rating Scale Self-assessment |
| MAR | Missing At Random |
| MCMC | Monte Carlo Markov Chain |
| MedDRA | Medical Dictionary for Regulatory Activities ICH |
| MMRM | Mixed-model repeated measures |
| MNAR | Missing Not At Random |
| OC | Observed Cases |
| PM | Poor metabolizer |
| PT | Preferred Term |
| QTc | QT corrected for heart rate |
| QTcB | QT corrected for heart rate by Bazett's formula |
| QTcF | QT corrected for heart rate by Fridericia's formula |
| QTcN | QT corrected for heart rate by FDA Neuropharmacological Division |
| | C 1 |

SDS

formula

Sheehan Disability Scale

#### Protocol 331-102-00058

SNRI Serotonin-noradrenaline reuptake inhibitor

SOC System Organ Class

SSRI Selective serotonin reuptake inhibitor TEAE Treatment-emergent adverse event

ULN Upper limit of normal

WHODD World Health Organization Drug Dictionary

## 1 Introduction

This statistical analysis plan documents in detail the statistical analysis methods planned for Trial 331-102-00058.

## 2 Trial Objectives

Primary endpoint: To assess the dosage and efficacy of brexpiprazole as adjunctive therapy vs placebo in combination with antidepressants (selective serotonin reuptake inhibitor [SSRI] or serotonin-noradrenaline reuptake inhibitor [SNRI]) in patients with major depressive disorder whose response to single-antidepressant therapy (SSRI or SNRI) was inadequate

Secondary endpoint: To assess the safety of brexpiprazole as adjunctive therapy vs placebo in combination with antidepressants (SSRI or SNRI) in patients with major depressive disorder whose response to single-antidepressant therapy (SSRI or SNRI) was inadequate

## 3 Trial Design

## 3.1 Type/Design of Trial

The trial is a multi-center, randomized, double-blind, placebo-controlled, parallel group-comparison trial to assess the efficacy and safety of brexpiprazole as adjunctive therapy in patients with major depressive disorder, who have received 1 to 3 adequate antidepressant drug treatments<sup>a</sup> for the current major depressive episode and have shown an inadequate response<sup>b</sup> to all of these treatments, and whose response during the antidepressant treatment period (Phase A) has also been inadequate.

The trial design is shown in Figure 3.1-1. The trial comprises a screening period, antidepressant treatment period (Phase A), double-blind period (Phase B) or antidepressant-responder treatment-continuation period (Phase A+), and post-treatment observation period.

With complete recovery from depressive symptoms and not the slightest improvement considered as 100% and 0%, respectively, patients carry out self-evaluations for improvement by antidepressant drug treatments used to date, from among 4 grades (< 25% Improvement, 25% to 49% Improvement, 50% to <75% Improvement, and  $\geq$  75% Improvement), with the evaluations corresponding to < 25% Improvement or 25% to 49% Improvement classified as inadequate response.

Patients who, among 1 to 3 adequate antidepressant drug treatments, have received treatment for

<sup>&</sup>lt;sup>a</sup>Definition of "adequate antidepressant drug treatment" is provided below.

Treatment with an antidepressant at an approved dose for at least 6 weeks (for combination therapy, treatment for at least 3 weeks)

<sup>&</sup>lt;sup>b</sup>Definition of "inadequate response" is provided below.

 $\geq$  6 weeks at least once (receiving only combination therapies for  $\geq$  3 weeks does not qualify) are eligible for selection.



Figure 3.1-1 Trial Design

#### 3.2 Trial Treatments

## 3.2.1 Antidepressant Treatment Period (Phase A)

#### 1) Drugs

Among commercially available SSRIs (fluvoxamine maleate, paroxetine hydrochloride hydrate, sertraline hydrochloride, and escitalopram oxalate) and SNRIs (milnacipran hydrochloride, duloxetine hydrochloride, and venlafaxine hydrochloride), one antidepressant that is different from the prior medications of antidepressant\*, plus the placebo tablet

## 2) Dose and regimen

In the antidepressant treatment period (Phase A), subjects will orally receive an antidepressant (SSRI or SNRI), which is different from the antidepressant prior

<sup>\*</sup>Antidepressant that meets the definition for "adequate antidepressant drug treatment" and has been taken at the time of informed consent.

medications, plus a placebo tablet once daily in a single-blind manner. The antidepressant (SSRI or SNRI) will be administered at the dose and regimen specified in the package insert, and the dose of the antidepressant will be progressively increased, within the approved dose range, to the maximum dose, as far as possible, in accordance with subject status; for the last 2 weeks of the 8-week period, dose and regimen will be fixed. A placebo tablet will be orally administered once daily. When an antidepressant cannot be administered at a fixed dose and regimen for the last 2 weeks of the 8-week antidepressant treatment period (Phase A) for tolerability-related reasons, the subject will be withdrawn from the trial.

3) Treatment period 8 weeks

## 3.2.2 Double-blind Period (Phase B)

At Week 8 of the antidepressant treatment period (Phase A), subjects who meet the criteria for proceeding to the double-blind period (Phase B) will proceed to the double-blind period (Phase B).

- 1) Drugs
- One commercially available antidepressant (SSRI or SNRI) used in the antidepressant treatment period (Phase A)
- Investigational medicinal product (IMP):
  - 1 mg/day group: brexpiprazole 1 mg tablet
  - 2 mg/day group: brexpiprazole 1 mg tablet (until observations, examinations, and assessments at Week 1) and brexpiprazole 2 mg tablet (after observations, examinations, and assessments at Week 1)
  - Placebo group: placebo tablet

#### 2) Dose and regimen

- Commercially available antidepressant (SSRI or SNRI):
  An antidepressant (SSRI or SNRI) used in the antidepressant treatment period (Phase A) will be continued with no changes from the final dose and regimen; no changes in dose, regimen, or drug will be allowed.
- IMP·
  - 1 mg/day group: One brexpiprazole 1 mg tablet will be orally administered once daily.
  - 2 mg/day group: Treatment will be started with brexpiprazole at 1 mg/day. One brexpiprazole 1 mg tablet will be orally administered once daily until observations, examinations, and assessments at Week 1. After the

- observations, examinations, and assessments at Week 1, one brexpiprazole 2 mg tablet will be orally administered once daily.
- Placebo group: One placebo tablet will be orally administered once daily.

## 3) Treatment period

6 weeks

## 3.2.3 Antidepressant-responder Treatment-continuation Period (Phase A+)

Antidepressant responders who do not meet the criteria for proceeding to the double-blind period (Phase B) based on the assessment at Week 8 of the antidepressant treatment period (Phase A) will proceed to the antidepressant-responder treatment-continuation period (Phase A+).

#### 1) Drugs

A commercially available antidepressant (SSRI or SNRI) used in the antidepressant treatment period (Phase A) plus the placebo tablet

#### 2) Dose and regimen

Subjects will receive an antidepressant (SSRI or SNRI) used in the antidepressant treatment period (Phase A) with no changes from the final dose and regimen, plus oral placebo (1 tablet) once daily in a single-blind manner.

## 3) Treatment period

6 weeks

#### 3.3 Trial Population

Adult patients with "major depressive disorder, single episode" or "major depressive disorder, recurrent episode" according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).

## 3.3.1 Number of Subjects and Trial Population

The trial will be conducted in patients 20 to < 65 years of age who have major depressive disorder (major depressive disorder, single episode; major depressive disorder, recurrent episode) according to the DSM-5 classification. After provision of informed consent, subjects considered eligible at the screening examination and at the examination performed at the initiation of the antidepressant treatment period (Phase A) will commence the antidepressant treatment period (Phase A) in which they will receive antidepressants different from their prior antidepressant medications (SSRI or SNRI) and

placebo tablets for 8 weeks in a single-blind manner. Subjects showing no response to the antidepressants during the antidepressant treatment period (Phase A) who meet the criteria for proceeding will proceed to the double-blind period (Phase B) to receive the IMP (brexpiprazole at 1 or 2 mg/day, or placebo) for 6 weeks in combination with the antidepressants used in the antidepressant treatment period (Phase A). The planned number of subjects proceeding to the double-blind period (Phase B) is set as follows: brexpiprazole 1 mg/day group: 240; brexpiprazole 2 mg/day group: 240; placebo group: 240; total: 720.

Subjects responding to antidepressants during the antidepressant treatment period (Phase A) and not meeting the criteria for proceeding to the double-blind period (Phase B) will not proceed to the double-blind period (Phase B) and will instead proceed to the antidepressant-responder treatment-continuation period (Phase A+), to receive 6-week treatment with placebo tablets in addition to the antidepressants (SSRI or SNRI) used in the antidepressant treatment period (Phase A), in a single-blind manner.

#### 3.4 Trial Visit Window

For all endpoints, acceptable windows for analysis are specified, and analysis should be based on the analysis time points regardless of time points recorded on the case report form.

Acceptable windows for analysis in the double-blind period (Phase B) are shown in Table 3.4-1. Day 1 is defined as the day when treatment with the IMP begins in the double-blind period. If multiple data exist within an acceptable window, the last data within the window will be used in analysis. Data obtained 7 days or later after the final dosing in the double-blind period will be excluded from the analysis.

| Table 3.4-1 Acceptable Windows for Analysis in the Double-blind Period (Phase B) | | |
|---|---|---|
| Week | Target Day | Trial Day Interval |
| Baseline | 1 | - 1 |
| Week 1 in the double-blind period | 7 | 2 - 10 |
| Week 2 in the double-blind period | 14 | 11 - 17 |
| Week 3 in the double-blind period | 21 | 18 - 24 |
| Week 4 in the double-blind period | 28 | 25 - 31 |
| Week 5 in the double-blind period | 35 | 32 - 38 |
| Week 6 in the double-blind period | 42 | 39 - 49 |

Acceptable windows for analysis in the antidepressant treatment period (Phase A) are shown in Table 3.4-2. Day 1 is defined as the day when treatment with the IMP begins in the antidepressant treatment period (Phase A). If multiple data exist within an acceptable window, the last data within the window will be used in analysis. Data obtained after

initiation of IMP treatment in the double-blind period (Phase B) or in the antidepressant-responder treatment-continuation period (Phase A+) and data obtained 7 days or later after the final dosing in the antidepressant treatment period (Phase A) will be excluded from the analysis.

| Table 3.4-2 Acceptable Windows for Analysis in the Antidepressant Treatment Period (Phase A) | | |
|---|---|---|
| Week | Target Day | Trial Day Interval |
| Baseline | 1 | - 1 |
| Week 1 in the antidepressant treatment period 7 2 - 10 | | |
| Week 2 in the antidepressant treatment period | 14 | 11 - 17 |
| Week 3 in the antidepressant treatment period 21 18 - 24 | | |
| Week 4 in the antidepressant treatment period 28 | | 25 - 31 |
| Week 5 in the antidepressant treatment period 35 32 - 38 | | 32 - 38 |
| Week 6 in the antidepressant treatment period 42 39 - 45 | | |
| Week 7 in the antidepressant treatment period 49 46 - 52 | | 46 - 52 |
| Week 8 in the antidepressant treatment period | 56 | 53 - 63 |

Acceptable windows for analysis in the antidepressant-responder treatment-continuation period (Phase A+) are the same as for the double-blind period (Phase B) (Table 3.4-1).

#### 3.5 Handling of Endpoints

## 3.5.1 Montgomery Asberg Depression Rating Scale (MADRS)

The MADRS total score will be the sum of scores for MADRS Items 1 through 10.

## 3.5.2 Clinical Global Impression – Improvement (CGI-I)

"0. Not assessed" will be handled as missing data.

#### 3.5.3 Clinical Global Impression - Severity of Illness (CGI-S)

"0. Not assessed" will be handled as missing data.

#### 3.5.4 Hamilton Rating Scale for Depression (HAM-D)

The HAM-D 17-item total score will be the sum of scores for HAM-D Items 1 through 17.

## 3.5.5 Sheehan Disability Scale (SDS)

The mean SDS score will be the mean of scores for 3 SDS items (work/school, social life, and family life/home responsibilities). In the case of a missing score for work/school, the mean of scores for the other 2 items will be handled as the mean SDS score.

# 3.5.6 Montgomery Asberg Depression Rating Scale Self-assessment (MADRS-S)

The MADRS-S total score will be the total score of MADRS-S Items 1 through 9.

#### 3.5.7 Drug-induced Extrapyramidal Symptoms Scale (DIEPSS)

The DIEPSS total score will be the sum of scores for DIEPSS items 1 through 8.

#### 3.5.8 Abnormal Involuntary Movement Scale (AIMS)

The AIMS total score will be the sum of scores for AIMS items 1 through 7.

## 4 Sample Size

In phase 3, double-blind, placebo-controlled, fixed dose trials of brexpiprazole (331-10-227, 331-10-228, and 331-13-214) conducted outside Japan, changes from baseline in MADRS total scores at Week 6 of the double-blind period (Phase B) have been analyzed by the Mixed-model Repeated Measure (MMRM) method (for 331-10-227 and 331-10-228, based on the results for efficacy from an analysis of subgroups meeting the inclusion criteria that had been revised in the middle of the trials), which demonstrated that the differences between the brexpiprazole groups (the 3 mg group in 331-10-227, and the 2 mg group in 331-10-228 and 331-13-214) and the placebo group were -1.9, -3.2, and -2.3, respectively, and that the standard deviations obtained from standard errors and numbers of subjects at Week 6 of the double-blind period (Phase B) were 7.2, 7.7, and 8.2, respectively. On the assumption that the difference in changes from baseline in MADRS total scores at Week 6 of the double-blind period (Phase B) is -2.4 for the brexpiprazole group compared with the placebo group with a standard deviation of 7.7. this trial will require 218 subjects per group to ensure a power of 90% in a two-sided test with a significance level of 0.05. We have decided that the planned number of subjects for randomization will be 240 per group, assuming that 7% of subjects will discontinue the trial during the double-blind period (Phase B) and some subjects will be excluded from analysis.

## 5 Statistical Analysis Datasets

## 5.1 Pharmacokinetic Analysis Set

The pharmacokinetic analysis set will comprise subjects who have been treated with brexpiprazole and for whom plasma brexpiprazole concentration data have been obtained.

## 5.2 Full Analysis Set

The full analysis set (FAS) will comprise subjects who, after randomization, have received at least 1 dose of the IMP in the double-blind period (Phase B), and from whom MADRS total scores have been obtained at baseline and at least 1 time point after initiation of the treatment

## 5.3 Safety Analysis Set

The safety analysis set will comprise subjects who, after randomization, have received at least 1 dose of the IMP in the double-blind period (Phase B).

## 5.4 Antidepressant Therapy Set

The antidepressant therapy (ADT) set will comprise subjects who have received at least 1 dose of the IMP in the antidepressant treatment period (Phase A).

## 5.5 Phase A+ Set

The Phase A+ set will comprise subjects who have received at least 1 dose of the IMP in the antidepressant-responder treatment-continuation period (Phase A+).

## 5.6 Handling of Missing Data

The primary analysis of the primary endpoint will be performed in the observed cases (OC) dataset by MMRM without data imputation for missing data under the missing at random (MAR) assumption. As a sensitivity analysis for the handling of missing data, placebo multiple imputation and tipping point analysis will be performed under the missing not at random (MNAR) assumption. Details are described in Section 8.1.2.

For efficacy and safety analyses, the last observation carried forward (LOCF) method (in which missing post-dose data are imputed by the last observed data after initiation of IMP treatment in the double-blind period) will be used as needed.

For pharmacokinetic analysis, no imputation will be performed for missing data.

## 6 Primary and Secondary Outcome Variables:

## 6.1 Primary Outcome Variables

Mean changes from baseline (Week 8 of the antidepressant treatment period [Phase A]) in MADRS total scores at Week 6 of the double-blind period (Phase B)

## 6.2 Secondary Outcome Variables

- MADRS response rate at Week 6 of the double-blind period (Phase B)
  The proportion of subjects in whom MADRS total scores at Week 6 of the double-blind period (Phase B) have been reduced by at least 50% from baseline (Week 8 of the antidepressant treatment period [Phase A])
- MADRS remission rate at Week 6 of the double-blind period (Phase B)
  The proportion of subjects in whom MADRS total scores at Week 6 of the double-blind period (Phase B) have been reduced by at least 50% from baseline (Week 8 of the antidepressant treatment period [Phase A]), with their MADRS total scores, at Week 6 of the double-blind period (Phase B), being ≤ 10
- CGI-I improvement rate at Week 6 of the double-blind period (Phase B)
  The proportion of subjects who score 1 or 2 on the CGI-I scale at Week 6 of the double-blind period (Phase B)
- Mean changes in CGI-S at Week 6 of the double-blind period (Phase B)
   Mean changes from baseline (Week 8 of the antidepressant treatment period [Phase A]) in CGI-S at Week 6 of the double-blind period (Phase B)
- Mean changes in HAM-D 17-item total scores at Week 6 of the double-blind period (Phase B)
   Mean changes from baseline (Week 8 of the antidepressant treatment period [Phase A]) in HAM-D 17-item total scores at Week 6 of the double-blind period (Phase B)
- Mean changes in mean SDS scores at Week 6 of the double-blind period (Phase B)
   Mean changes from baseline (Week 8 of the antidepressant treatment period [Phase A]) in mean SDS scores at Week 6 of the double-blind period (Phase B)
- Mean changes in MADRS-S total scores at Week 6 of the double-blind period (Phase B)
   Mean changes from baseline (Week 8 of the antidepressant treatment period [Phase A]) in MADRS-S total scores at Week 6 of the double-blind period (Phase B)

## 7 Disposition and Demographic Analysis

## 7.1 Subject Disposition

Numbers and proportions of subjects from whom informed consent was obtained, those who received trial treatment in the antidepressant treatment period (Phase A), those who completed the antidepressant treatment period (Phase A), those who discontinued treatment in the antidepressant treatment period (Phase A), those who discontinued treatment in the antidepressant treatment period (Phase A) by reason, and those who were included in the ADT set will be summarized overall and for each requisite concomitant medication.

Numbers and proportions of randomized subjects in the double-blind period (Phase B), those who received trial treatment in the double-blind period (Phase B), those who

completed the double-blind period (Phase B), those who discontinued treatment in the double-blind period (Phase B), those who discontinued treatment in the double-blind period (Phase B) by reason, and those who were included in each analysis set will be summarized overall, for each treatment group, and for the overall brexpiprazole group. Similar summarization will be performed for each requisite concomitant medication.

Numbers and proportions of subjects who received trial treatment in the antidepressant-responder treatment-continuation period (Phase A+), those who completed the antidepressant-responder treatment-continuation period (Phase A+), those who discontinued treatment in the antidepressant-responder treatment-continuation period (Phase A+), those who discontinued treatment in the antidepressant-responder treatment-continuation period (Phase A+) by reason, and those who were included in the Phase A+ set will be summarized overall and for each requisite concomitant medication.

Numbers and proportions of subjects who completed the double-blind period (Phase B) will be summarized by each period (days) (1-7, 8-14, 15-21, 22-28, 29-35, 36-42, and > 42) overall, for each treatment group, and for the overall brexpiprazole group.

#### 7.2 Demographic and Baseline Characteristics

Descriptive statistics (mean, standard deviation, minimum, median, maximum; hereinafter the same applies) of age, height, body weight, waist circumference, and body mass index (BMI) and frequency distribution of age ( $<55, \ge 55$ ), sex, race, ethnicity, country where trial is conducted, medical history, complications, and CYP2D6 phenotype will be determined overall, for each treatment group, and for the overall brexpiprazole group in each analysis set in the double-blind period (Phase B). Similar summarization will be performed for each requisite concomitant medication in the safety analysis set and the FAS.

Similar summarization (but not for CYP2D6 phenotype) will be performed overall and for each requisite concomitant medication in the ADT set and the Phase A+ set.

Baseline data in each period will be used for body weight, waist circumference, and BMI.

#### 7.3 Baseline Disease Evaluation

Descriptive statistics of the duration (months) of the current major depressive episode, age at initial onset, duration (months) of major depressive episode from initial onset, MADRS total score, HAM-D 17 total score, and CGI-S and frequency distribution of DSM-5-based diagnosis (single, recurrent), severity (mild, moderate, severe), specific terms ("not applicable," "applicable," and disposition of each specific term), frequency of major depressive episodes  $(1, 2, 3, 4, \ge 5)$ , frequency of appropriate antidepressant drug

treatments of the current major depressive episode (1, 2, 3) will be determined overall, for each treatment group, and for the overall brexpiprazole group in the safety analysis set and the FAS. Similar summarization will be performed for each requisite concomitant medication.

Similar summarization will be performed overall and for each requisite concomitant medication in the ADT set and the Phase A+ set.

For the double-blind period (Phase B), values at baseline (8 weeks after the antidepressant treatment period [Phase A]) and at the start of the antidepressant treatment period (Phase A) will be used for MADRS total score, HAM-D 17 total score, and CGI-S. For the ADT set and the Phase A+ set, values at the start of the antidepressant treatment period (Phase A) will be used for those scores.

The duration of the current major depressive episode and the duration of major depressive episode from initial onset will be calculated using the following formula: duration (months) = (date of subject demographic evaluation – date of onset + 1) / 30. Any unknown month or day of onset will be replaced with June or 15, respectively.

#### 7.4 Treatment Compliance

Treatment compliance (number of days when the subject actually received the IMP/number of days for which the IMP was prescribed) in the double-blind period (Phase B) will be grouped into < 70%,  $\ge 70\%$  to < 80%,  $\ge 80\%$  to < 90%, and  $\ge 90\%$ , and its frequency distribution will be determined overall, for each treatment group, and for the overall brexpiprazole group in the FAS.

#### 7.5 Prior and Concomitant Medications

Numbers and proportions of subjects who used medications before the antidepressant treatment period (Phase A), during the antidepressant treatment period (Phase A) and the double-blind period (Phase B), and after the double-blind period (Phase B) will be determined by drug class and preferred term of the World Health Organization Drug Dictionary (WHODD) version Global B3 March 2018 overall, for each treatment group, and for the overall brexpiprazole group in the safety analysis set.

Medications used in the antidepressant treatment period (Phase A) will be similarly summarized overall and for each requisite concomitant medication in the ADT set. Medications used in the antidepressant-responder treatment-continuation period (Phase A+) will also be similarly summarized overall and for each requisite concomitant medication in the Phase A+ set.

Similar summarization will be performed for antipsychotics.

#### 7.6 Protocol Deviations

In randomized subjects, numbers and proportions of subjects with major deviations from the protocol will be determined for each deviation category (treatment-related deviations, eligibility-related deviations, a failure to discontinue the trial when the subject meets the withdrawal criteria, procedure-related deviations that affect evaluation of the primary endpoint, use of prohibited medications, and overall) and each trial site, overall, for each treatment group, and for the overall brexpiprazole group.

In non-randomized subjects, similar summarization will be performed overall and for each requisite concomitant medication.

## 8 Efficacy Analysis

Efficacy analysis in the double-blind period (Phase B) will be performed using the FAS. Unless otherwise stated, the efficacy analysis described in this section relates only to the double-blind period (phase B).

#### 8.1 Primary Efficacy Endpoint

The primary endpoint is mean changes from baseline (Week 8 of the antidepressant treatment period [Phase A]) in MADRS total scores at Week 6 of the double-blind period (Phase B).

## 8.1.1 Primary Efficacy Analysis

For the primary analysis, MMRM analysis will be performed using the OC data set in the FAS. The statistical hypotheses will be tested, based on differences in least square means between each brexpiprazole group and the placebo group, which are calculated by MMRM. To adjust for multiplicity of tests, due to there being 2 comparisons with the placebo group for each of the brexpiprazole groups, a fixed-sequence approach will be used to control overall type 1 error rates. Comparison between the brexpiprazole 2 mg/day group and placebo group will be performed first; only when significance is observed at a two-sided significance level of 5%, will comparison between the brexpiprazole 1 mg/day group and placebo group be performed at a two-sided significance level of 5%.

The MMRM will include treatment group (brexpiprazole 1 mg/day group, brexpiprazole 2 mg/day group, and placebo group), time point (double-blind period [Phase B] Weeks 1, 2, 3, 4, 5, and 6), and interaction between treatment group and time point as factors, and baseline and interaction between baseline and time point as covariates. Unstructured error variance-covariance structure will be assumed. For a degree-of-freedom approximation,

the Kenward-Roger method will be used. If any problems in convergence status arise in the estimation of variance components, heterogeneous Toeplitz, heterogeneous autoregressive of order 1, and heterogeneous compound symmetry, which are error variance-covariance structures, will be applied in this order, and the first structure that achieves convergence will be used in the primary analysis. If anything other than an unstructured variance-covariance structure is selected, a sandwich estimator for standard errors will be used.

For each time point, least square means of each treatment group and differences in least square means between each brexpiprazole group and the placebo group, as well as the two-sided 95% confidence intervals (CIs) will be determined.

## 8.1.2 Sensitivity Analyses

## 8.1.2.1 Sensitivity Analysis for Handling of Missing Data

As a sensitivity analysis for handling of missing data, placebo multiple imputation and tipping point analysis on MNAR assumption will be performed using a pattern-mixture model with multiple imputation.

Multiple imputation analysis will be performed according to the following procedure. The number of imputations will be 100.

- 1) The Markov Chain Monte Carlo (MCMC) method will be used to impute intermittent missing data to produce a monotone missing data pattern.
- 2) The monotone regression method will be used to impute monotone missing data.
- 3) The same MMRM as that of the primary efficacy analysis will be used to analyze the multiple-imputed datasets.
- 4) The MIANALYZE procedure will be used to integrate the analysis results of the multiple-imputed datasets, and the estimate of the difference between each brexpiprazole group and the placebo group at Week 6 in the double-blind period (Phase B) and its 95% CI and p-value will be determined.

In placebo multiple imputation, for discontinued subjects in each brexpiprazole group, MNAR will be assumed for missing data after discontinuation and an imputation model based on the placebo group will be used in imputation.

In tipping point analysis, for subjects in each brexpiprazole group who discontinued treatment for any of the following reasons, MNAR will be assumed for missing data after discontinuation.

- Withdrawal for any reason
- Withdrawal due to AEs, a lack of efficacy, or consent withdrawal
- Withdrawal due to AEs or a lack of efficacy

For subjects in each brexpiprazole group who discontinued treatment for reasons assumed as MNAR, the MAR assumption will be used to impute post-discontinuation missing data, add  $\Delta$  (intergroup differences in MMRM of the primary efficacy analysis) × k% to the imputed value, and increase k until a statistically significant conclusion is reversed (p > 0.05).

## 8.1.2.2 Sensitivity Analysis for Normality Assumption

As a sensitivity analysis for normality assumption, multiple imputation under the MAR assumption will be performed, and the Wilcoxon rank sum test will be used to compare each brexpiprazole group and the placebo group for each time point, and the Hodges-Lehmann estimator of the intergroup difference will be determined. A robust regression analysis with treatment group as a factor and baseline as a covariate will also be performed for each time point. Similar analysis without multiple imputation will also be performed.

## 8.1.3 Technical Computational Details for Primary Efficacy Analysis

The SAS code for the MIXED procedure to perform the primary efficacy MMRM analysis is shown below.

```
proc mixed;
```

run;

```
class treatment visit subjid;
model change=treatment visit baseline treatment*visit baseline*visit / ddfm=kr;
repeated visit /type=un subject=subjid;
lsmeans treament*visit / diff cl;
ods output diffs=diffs lsmeans=lsmeans;
```

## 8.2 Secondary Efficacy Analyses

- MADRS response rate at Week 6 of the double-blind period (Phase B)
- MADRS remission rate at Week 6 of the double-blind period (Phase B)
- CGI-I improvement rate at Week 6 of the double-blind period (Phase B)

For the MADRS response rate, a  $\chi^2$  test will be performed for between-treatment-group comparison using the LOCF data set. Differences in the response rates between each of the brexpiprazole groups and the placebo group, and the two-sided 95% CIs (Wald confidence interval) will be determined. For MADRS remission rate and CGI-I

improvement rate, the same analysis employed for the MADRS response rate will be used. The same analysis will be performed on the OC dataset.

- Mean changes from baseline (Week 8 of the antidepressant treatment period [Phase A]) in HAM-D 17-item total scores at Week 6 of the double-blind period (Phase B) Using the LOCF data set, analysis will be performed by ANCOVA model with treatment group as a factor and baseline as a covariate. Least square means of each treatment group and differences in least square means between each brexpiprazole group and the placebo group, as well as the two-sided 95% CIs will be determined. The same analysis will be performed on the OC dataset.
- Mean changes from baseline (Week 8 of the antidepressant treatment period [Phase A]) in CGI-S at Week 6 of the double-blind period (Phase B)
- Mean changes from baseline (Week 8 of the antidepressant treatment period [Phase A]) in mean SDS scores at Week 6 of the double-blind period (Phase B)
- Mean changes from baseline (Week 8 of the antidepressant treatment period [Phase A]) in MADRS-S total scores at Week 6 of the double-blind period (Phase B)

As performed for the primary endpoint, MMRM analysis will be performed. Each item on the SDS (work/school, social life, and family life/home responsibilities) will also be analyzed in the same manner.

## 8.3 Subgroup Analyses

For the change from baseline (Week 8 of the antidepressant treatment period [Phase A]) in MADRS total score, the same MMRM analysis as that of the primary endpoint will be performed for each of the following subgroups.

For CYP2D6 phenotype, all subjects in the placebo group will be included in each subgroup.

- Requisite concomitant medication (duloxetine, escitalopram, fluvoxamine, milnacipran, paroxetine, sertraline, venlafaxine)
- Sex (male, female)
- Age  $(< 55, \ge 55)$
- Number of adequate antidepressant drug treatments (1, 2, 3)
- DSM-5 diagnosis (single episode, recurrent episode)
- Frequency of major depressive episodes  $(1, 2, \ge 3)$
- Duration (in months) of the current episode (≤ median, > median)
- Baseline MADRS total score (≤ median, > median)

- Concomitant use of ultrashort-acting sedative-hypnotic drugs in the double-blind period (Phase B) (yes or no)
- Body weight (≤ median, > median)
- BMI ( $\leq$  median, > median)
- CYP2D6 phenotype (IM, EM)
- Impact of COVID-19 pandemic (subjects from whom consent was obtained before 07 Apr 2020, those from whom consent was obtained on or after 07 Apr 2020)

## 8.4 Exploratory or Other Analyses

The Cochran Mantel Haenszel (CMH) Row Mean Scores test of CGI-I scores will be performed on the LOCF dataset to compare each brexpiprazole group and the placebo group. The mean in each treatment group and the mean difference between each brexpiprazole group and the placebo group with their two-sided 95% CIs will be determined. The same analysis will be performed on the OC dataset.

The MADRS total score, CGI-I, CGI-S, mean SDS score and the score of each item, and MADRS-S total score at each time point in the double-blind period (Phase B) will be analyzed in the FAS in the same manner as for the primary and secondary endpoints. Descriptive statistics or frequency distribution of actual measurements and changes from baseline at each time point will be calculated by treatment group.

For MADRS total score, HAM-D 17-item total score, CGI-S, mean SDS score and the score of each item, and MADRS-S total score in the antidepressant treatment period (Phase A), descriptive statistics of actual measurements and changes from baseline (before the start of the antidepressant treatment period [Phase A]) will be calculated overall and for each requisite concomitant medication in the ADT set.

For MADRS total score, HAM-D 17-item total score, CGI-S, mean SDS score and the score of each item, and MADRS-S total score in the antidepressant treatment period (Phase A) and the antidepressant-responder treatment-continuation period (Phase A+), descriptive statistics of actual measurements and changes from baseline (before the start of the antidepressant treatment period [Phase A]) will be calculated overall and for each requisite concomitant medication in the Phase A+ set.

## 9 Safety Analyses

Safety analysis for the double-blind period (Phase B) will be performed using the safety analysis set. Unless otherwise stated, the safety analysis described in this section relates only to the double-blind period (phase B).

## 9.1 Extent of Exposure

Frequency distribution of the duration (in days) of treatment with the IMP in the double-blind period (Phase B) (1-7, 8-14, 15-21, 22-28, 29-35, 36-42, and > 42) will be determined by treatment group and for the overall brexpiprazole group. Similar summarization will be performed for each requisite concomitant medication subgroup.

Frequency distribution of the duration (in days) of treatment with a requisite concomitant medication in the double-blind period (Phase B) (1-7, 8-14, 15-21, 22-28, 29-35, 36-42, and > 42) will be determined by treatment group and for the overall brexpiprazole group.

Descriptive statistics of the mean daily dose of each requisite concomitant medication in the double-blind period (Phase B) will be calculated by treatment group and for the overall brexpiprazole group.

Frequency distribution of the duration (in days) of treatment with a requisite concomitant medication in the antidepressant treatment period (Phase A) (1-7, 8-14, 15-21, 22-28, 29-35, 36-42, 43-49, 50-56, and > 56) will be determined overall and for each requisite concomitant medication in the ADT set.

Frequency distribution of the duration (in days) of treatment with a requisite concomitant medication in the antidepressant-responder treatment-continuation period (Phase A+) (1-7, 8-14, 15-21, 22-28, 29-35, 36-42, and > 42) will be determined overall and for each requisite concomitant medication in the Phase A+ set.

#### 9.2 Adverse Events

All adverse events (AEs) will be coded by Medical Dictionary for Regulatory Activities (MedDRA) (Ver. 24.0) System Organ Class (SOC) and Preferred Term (PT). Numbers and proportions of subjects with the following AEs will be summarized by SOC and PT by treatment group and for the overall brexpiprazole group. If an AE occurs more than once in the same subject, the severest event will be used in summarization.

- Adverse events occurring after initiation of IMP administration in the double-blind period (Phase B) (treatment-emergent adverse events [TEAEs])
- TEAEs by severity
- TEAEs with an outcome of death
- Serious TEAEs
- TEAEs leading to discontinuation of the IMP
- TEAEs occurring in  $\geq$  2% of subjects in any brexpiprazole group and more frequently than in the placebo group

• TEAEs by date of initial onset (1-7, 8-14, 15-21, 22-28, 29-35, 36-42, > 42, post-trial treatment)

TEAEs potentially causally related to the IMP will also be summarized in the same manner.

#### 9.2.1 Adverse Events of Interest

Each adverse event of interest is defined in Appendix 4. Numbers and proportions of subjects with the following AEs of interest will be summarized by SOC and PT by treatment group and for the overall brexpiprazole group.

- Extrapyramidal AEs
- Neuroleptic malignant syndrome-related AEs
- Rhabdomyolysis
- Seizure-related AEs
- Orthostatic disorder-related AEs
- Suicide/suicide attempt-related AEs
- Oversedation-related AEs
- Hypersensitive symptom-related AEs
- Venous thrombosis
- Blood disorder-related AEs
- Glucose metabolism-related AEs
- Lipid metabolism-related AEs
- Body weight-related AEs
- QT interval prolongation-related AEs
- Manic switch-related AEs
- Prolactin increase-related AEs

## 9.2.2 Subgroup Analysis of Adverse Events

Numbers and proportions of subjects with TEAEs will be summarized by SOC and PT by treatment group and for the overall brexpiprazole group in each of the following subgroups:

- Requisite concomitant medication (duloxetine, escitalopram, fluvoxamine, milnacipran, paroxetine, sertraline, venlafaxine)
- Sex (male, female)
- Age  $(< 55, \ge 55)$
- CYP2D6 phenotype (IM, EM, PM, Unknown)

• Impact of COVID-19 pandemic (subjects from whom consent was obtained before 07 Apr 2020, those from whom consent was obtained on or after 07 Apr 2020)

# 9.2.3 Adverse Events in the Antidepressant Treatment Period (Phase A) and the Antidepressant-responder Treatment-continuation Period (Phase A+)

Numbers and proportions of subjects who experienced AEs in the antidepressant treatment period (Phase A) will be summarized by SOC and PT overall and for each requisite concomitant medication in the ADT set.

Numbers and proportions of subjects who experienced AEs in the antidepressant-responder treatment-continuation period (Phase A+) will be summarized by SOC and PT overall and for each requisite concomitant medication in the Phase A+ set.

## 9.3 Clinical Laboratory Data

For each quantitative laboratory parameter, descriptive statistics of actual measurements and changes from baseline at each time point and the last time point will be calculated for each treatment group and for the overall brexpiprazole group.

For each quantitative laboratory parameter, actual measurements will be classified as "lower than the lower limit of the reference range," "within the reference range," and "higher than the upper limit of the reference range" using the reference range specified by the central laboratory, and a shift table from baseline will be produced for each treatment group and for the overall brexpiprazole group.

For each qualitative laboratory parameter, a shift table from baseline will be produced for each treatment group and for the overall brexpiprazole group.

Numbers and proportions of subjects with laboratory test values not meeting the criteria for potentially clinically significant laboratory test values (Appendix 2) at baseline and meeting the criteria after treatment will be determined for each treatment group and for the overall brexpiprazole group. A listing of these subjects will be provided.

Numbers and proportions of subjects with postdose values of alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin (TBL) meeting Hy's Law criteria (ALT or AST  $\geq$  3 × the upper limit of normal [ULN] and TBL  $\geq$  2 × ULN) will be determined for each treatment group and for the overall brexpiprazole group. A listing of these subjects will be provided.

Numbers and proportions of subjects with a prolactin value not meeting the criteria of  $> 1 \times ULN$ ,  $> 2 \times ULN$ , or  $> 3 \times ULN$  at baseline and meeting the criteria after treatment

will be determined by sex for each treatment group and for the overall brexpiprazole group. A listing of these subjects will be provided.

Numbers and proportions of subjects with postdose values of fasting low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, triglyceride, and blood glucose meeting the criteria for changes in glucose and lipid metabolism-related parameters (Table 9.3-1) will be determined by baseline value for each treatment group and for the overall brexpiprazole group. A listing of these subjects will be provided.

| Table 9.3-1 Changes in Glucose and Lipid Metabolism-related | | |
|---|---|---|
| Parameters | | |
| LAB PARAMETER | BASELINE | ANYTIME POST BASELINE |
| LDL Cholesterol, Fasting | Borderline 100-<160 | High >=160 |
| (mg/dL) | Normal/Borderline < 160 | High >=160 |
| | Normal <100 | Borderline/High >=100 |
| | Any Value | Increased >=30 |
| HDL Cholesterol, Fasting | Normal >=40 | Low <40 |
| (mg/dL) | Any Value | Decreased >=20 |
| Triglycerides, Fasting | Normal <150 | High 200-<500 |
| (mg/dL) | Borderline 150-<200 | High 200-<500 |
| | Normal/Borderline <200 | High 200-<500 |
| | Normal <150 | Borderline/High/Very High >=150 |
| | Normal/Borderline/high <500 | Very High >=500 |
| | Any Value | Increased >=50 |
| Glucose Fasting, Serum | Normal <100 | High >=126 |
| (mg/dL) | Impaired 100-<126 | High >=126 |
| | Normal/Impaired <126 | High >=126 |
| | Any Value | Increased >=10 |

Numbers and proportions of subjects not meeting the metabolic syndrome criteria (Table 9.3-2) at baseline and meeting the criteria after treatment will be determined for each treatment group and for the overall brexpiprazole group. A listing of these subjects will be provided.

| Table 9.3-2 Metabolic Syndrome Criteria | |
|---|---|
| Description | Metabolic Syndrome Criteria (Health, Labour and Welfare Ministry of Japan) |
| Central obesity | Waist Circumference ≥85 cm (Male), ≥90 cm (Female) |
| Dyslipidemia | Triglycerides, Fasting ≥150 mg/dL and/or HDL, Fasting <40 mg/dL |
| Supine blood pressure | Systolic ≥130 mmHg and/or Diastolic ≥85 mmHg |
| Glucose fasting, serum | $\geq$ 110 mg/dL |
| Metabolic syndrome | met central obesity criteria and 2 of 3 other criteria at a visit |

For each quantitative laboratory parameter in the antidepressant treatment period (Phase A), descriptive statistics of actual measurements and changes from baseline (before the

start of the antidepressant treatment period [Phase A]) at each time point and the last assessment time point will be calculated overall and for each requisite concomitant medication in the ADT set. A listing of subjects with laboratory test values meeting the criteria for potentially clinically significant laboratory test values (Appendix 2) will be provided.

For each quantitative laboratory parameter in the antidepressant treatment period (Phase A) and the antidepressant-responder treatment-continuation period (Phase A+), descriptive statistics of actual measurements and changes from baseline (before the start of the antidepressant treatment period [Phase A]) at each time point and the last assessment time point will be calculated overall and for each requisite concomitant medication in the Phase A+ set. A listing of subjects with laboratory test values meeting the criteria for potentially clinically significant laboratory test values (Appendix 2) will be provided.

## 9.4 Vital Sign Data

For each vital sign parameter (by position for blood pressure and pulse rate), descriptive statistics of actual measurements and changes from baseline at each time point and the last assessment time point will be calculated for each treatment group and for the overall brexpiprazole group.

Numbers and proportions of subjects with vital signs meeting the criteria for potentially clinically significant vital signs (Appendix 1) will be determined for each treatment group and for the overall brexpiprazole group. A listing of these subjects will be provided.

For each vital sign parameter in the antidepressant treatment period (Phase A), descriptive statistics of actual measurements and changes from baseline (before the start of the antidepressant treatment period [Phase A]) at each time point and the last assessment time point will be calculated overall and for each requisite concomitant medication in the ADT set. A listing of subjects with vital signs meeting the criteria for potentially clinically significant vital signs (Appendix 1) will be provided.

For each vital sign parameter in the antidepressant treatment period (Phase A) and the antidepressant-responder treatment-continuation period (Phase A+), descriptive statistics of actual measurements and changes from baseline (before the start of the antidepressant treatment period [Phase A]) at each time point and the last assessment time point will be calculated overall and for each requisite concomitant medication in the Phase A+ set. A listing of subjects with vital signs meeting the criteria for potentially clinically significant vital signs (Appendix 1) will be provided.

## 9.5 Physical Examination Data

Physical examination data will be provided in a listing.

## 9.6 Electrocardiogram Data

For heart rate, PR interval, RR interval, QRS interval, QT interval, and QT corrected for heart rate (QTc), descriptive statistics of actual measurements and changes from baseline at each time point and the last time point will be calculated for each treatment group and for the overall brexpiprazole group.

A shift table from baseline for normal/abnormal 12-lead electrocardiogram (ECG) (evaluated at the trial site) will be produced for each treatment group and for the overall brexpiprazole group.

Numbers and proportions of subjects with actual measurements of QTc (QTcF, QTcB, QTcN) not meeting the criteria of > 450 msec, > 480 msec, and > 500 msec at baseline and meeting the criteria after treatment will be determined for each treatment group and for the overall brexpiprazole group. Numbers and proportions of subjects with actual measurements of > 450 msec with a % change from baseline of > 10% will be determined for each treatment group and for the overall brexpiprazole group.

Numbers and proportions of subjects with ECG results meeting the criteria for potentially clinically significant ECG data (Appendix 3) will be determined for each treatment group and for the overall brexpiprazole group. A listing of these subjects will be provided.

For each ECG parameter in the antidepressant treatment period (Phase A), descriptive statistics of actual measurements and changes from baseline (before the start of the antidepressant treatment period [Phase A]) at each time point and the last assessment time point will be calculated overall and for each requisite concomitant medication in the ADT set. A listing of subjects with ECG results meeting the criteria for potentially clinically significant ECG data (Appendix 3) will be provided.

For each ECG parameter in the antidepressant treatment period (Phase A) and the antidepressant-responder treatment-continuation period (Phase A+), descriptive statistics of actual measurements and changes from baseline (before the start of the antidepressant treatment period [Phase A]) at each time point and the last assessment time point will be calculated overall and for each requisite concomitant medication in the Phase A+ set. A listing of subjects with ECG results meeting the criteria for potentially clinically significant ECG data (Appendix 3) will be provided.

## 9.7 Other Safety Data

## 9.7.1 Body Weight, BMI, and Waist Circumference

For body weight, BMI, and waist circumference, descriptive statistics of actual measurements and changes from baseline at each time point and the last assessment time point will be calculated for each treatment group and for the overall brexpiprazole group.

In addition, analysis will be performed by the ANCOVA model with treatment group as a factor and baseline as a covariate. Least square means of each treatment group and differences in least square means between each brexpiprazole group and the placebo group, as well as the two-sided 95% CIs will be determined.

Numbers and proportions of subjects with results meeting the criteria for potentially clinically significant body weight gain or loss (Appendix 1) will be determined for each treatment group and for the overall brexpiprazole group. Body weight data will also be analyzed by baseline BMI category ( $< 18.5, \ge 18.5$  to  $< 25, \ge 25$  to  $< 30, \ge 30$ ) in a similar manner. A listing of subjects with results meeting the criteria for potentially clinically significant body weight gain or loss (Appendix 1) will be provided.

For body weight, BMI, and waist circumference in the antidepressant treatment period (Phase A), descriptive statistics of actual measurements and changes from baseline (before the start of the antidepressant treatment period [Phase A]) at each time point and the last assessment time point will be calculated overall and for each requisite concomitant medication in the ADT set. A listing of subjects with results meeting the criteria for potentially clinically significant body weight gain or loss (Appendix 1) will be provided.

For body weight, BMI, and waist circumference in the antidepressant treatment period (Phase A) and the antidepressant-responder treatment-continuation period (Phase A+), descriptive statistics of actual measurements and changes from baseline (before the start of the antidepressant treatment period [Phase A]) at each time point and the last assessment time point will be calculated overall and for each requisite concomitant medication in the Phase A+ set. A listing of subjects with results meeting the criteria for potentially clinically significant body weight gain or loss (Appendix 1) will be provided.

## 9.7.2 DIEPSS, AIMS, and Barnes Akathisia Rating Scale (BARS)

For DIEPSS total score (total of scores for items 1 through 8) and score for each DIEPSS item, AIMS total score (total of scores for items 1 through 7) and score for each of the items 8 through 10, and BARS, descriptive statistics of actual measurements and changes from baseline at each time point and the last assessment time point and the worst

postdose measurement and its change from baseline will be calculated for each treatment group and for the overall brexpiprazole group.

In addition, analysis will be performed by the ANCOVA model with treatment group as a factor and baseline as a covariate. Least square means of each treatment group and differences in least square means between each brexpiprazole group and the placebo group, as well as the two-sided 95% CIs will be determined.

For DIEPSS total score (total of scores for items 1 through 8) and score for each DIEPSS item, AIMS total score (total of scores for items 1 through 7) and score for each of the items 8 through 10, and BARS in the antidepressant-responder treatment-continuation period (Phase A+), descriptive statistics of actual measurements and changes from baseline (before the start of the antidepressant-responder treatment-continuation period [Phase A+]) at each time point and the last assessment time point will be calculated overall and for each requisite concomitant medication in the Phase A+ set.

## 9.7.3 Columbia-Suicide Severity Rating Scale (C-SSRS)

Numbers and proportions of subjects for each C-SSRS item (suicidality, suicidal ideation, suicidal behavior, completed suicide, emergence of suicidal ideation, emergence of serious suicidal ideation, worsening of suicidal ideation, and emergence of suicidal behavior) at each time point and in the overall period after initiation of IMP treatment in the double-blind period (including the post-treatment observation period, at discontinuation, and unscheduled visits) will be determined for each treatment group and for the overall brexpiprazole group. A listing of subjects with emergence of suicidal ideation, emergence of serious suicidal ideation, worsening of suicidal ideation, and emergence of suicidal behavior will be provided. Items of suicidal ideation and suicidal behavior will also be summarized in the same manner.

- Suicidality: "Yes" for any item of suicidal ideation or suicidal behavior
- Suicidal ideation: "Yes" for any item of suicidal ideation
- Suicidal behavior: "Yes" for any item of suicidal behavior
- Emergence of suicidal ideation: Change from "No" at baseline to "Yes" after baseline for suicidal ideation
- Emergence of serious suicidal ideation: Change from "No" at baseline to "Yes" with Grade 4 or 5 after baseline for suicidal ideation
- Worsening of suicidal ideation: Increase in the grade of suicidal ideation from baseline
- Emergence of suicidal behavior: Change from "No" at baseline to "Yes" after baseline for suicidal behavior

Items of suicidal ideation and suicidal behavior in the antidepressant treatment period (Phase A) will also be summarized in the ADT set.

Items of suicidal ideation and suicidal behavior in the antidepressant-responder treatment-continuation period (Phase A+) will also be summarized in the Phase A+ set.

## 10 Pharmacokinetic Analyses

Pharmacokinetic analysis will be performed on the pharmacokinetic analysis set.

Descriptive statistics of plasma brexpiprazole concentrations at time points (0-6, 6-12, 12-18, 18-24, 24-30, and > 30 hours) after the most recent dosing as well as trough brexpiprazole concentrations (20-28 hours after the most recent dosing) and plasma brexpiprazole concentrations at all time points will be calculated by treatment group. The descriptive statistics will also be calculated by CYP2D6 phenotype (EM, IM, PM, and Unknown) in each treatment group and by requisite concomitant medication in each treatment group in the same manner.

The mean plasma brexpiprazole concentration over time and individual values at each time point after the most recent dosing will be plotted by treatment group. Plotted diagrams by CYP2D6 phenotype in each treatment group and by requisite concomitant medication in each treatment group will also be provided in the same manner.

Scatter plots of plasma brexpiprazole concentrations over time will be provided by treatment group. Scatter plots by CYP2D6 phenotype in each treatment group and by requisite concomitant medication in each treatment group will also be provided in the same manner

Plasma brexpiprazole concentrations below the lower limit of quantitation will be handled as 0 (ng/mL) when their descriptive statistics are calculated and when plotted diagrams and scatter plots are created.

## 11 Pharmacodynamic Analyses

Not applicable.

## 12 Pharmacogenomic Analyses

CYP2D6 genotype (phenotype) will be tabulated as specified in Section 7.2 Demographic and Baseline Characteristics. CYP2D6 phenotype will also be summarized in subgroup efficacy and safety analyses.

## 13 Interim Analysis

No interim analyses are planned.

## 14 Changes in the Planned Analyses

- The following changes were made to categorical analyses of QTc:
   Only subjects with postdose QTc meeting the criteria will be summarized, instead of summarization at all time points.
  - Only subjects with QTc not meeting the criteria at baseline and meeting the criteria after baseline will be summarized.
- It has been decided that CYP2D6 phenotype will be tabulated as specified in Section 7.2 Demographic and Baseline Characteristics. CYP2D6 phenotype will also be summarized in subgroup efficacy and safety analyses.
- The original plan of using the LOCF dataset in ANCOVA of safety endpoints was changed as follows: Measurements at each time point and at the last assessment time point and, as necessary, the worst postdose measurement will be included in the analysis.
- The original plan of calculating descriptive statistics of plasma brexpiprazole
  concentrations by treatment group in pharmacokinetic analysis was changed as
  follows: Descriptive statistics of plasma brexpiprazole concentrations at each time
  point after the most recent dosing, trough concentrations, and plasma drug
  concentrations at all time points will be calculated by treatment group, by CYP2D6
  phenotype in each treatment group, and by requisite concomitant medication in each
  treatment group.

#### 15 References

Not applicable.

# Appendix 1 Criteria for Identifying Vital Signs and Weight of Potential Clinical Relevance

| Variable | Criterion Value <sup>a</sup> | Change Relative to Baseline <sup>a</sup> |
|---|---|---|
| Pulse Rate | > 120 bpm | ≥ 15 bpm increase |
| Fulse Kate | < 50 bpm | ≥ 15 bpm decrease |
| Systolic Blood Pressure | > 180 mmHg | ≥ 20 mmHg increase |
| Systolic Blood Flessule | < 90 mmHg | ≥ 20 mmHg decrease |
| Diastolic Blood Pressure | > 105 mmHg | ≥ 15 mmHg increase |
| Diastolic Blood Plessure | < 50 mmHg | ≥ 15 mmHg decrease |
| Orthostatic Hypotension | ≥ 20 mmHg decrease in systolic blood<br>pressure and a ≥ 25 bpm increase in<br>pulse rate from supine to<br>sitting/standing | Not Applicable |
| Weight | - | ≥ 7% increase<br>≥ 7% decrease |

<sup>&</sup>lt;sup>a</sup>In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.

Appendix 2 Criteria for Identifying Laboratory Values of Potential Clinical Relevance

| Laboratory Tests | Criteria |
|---|---|
| Chemistry | |
| AST (SGOT) | ≥ 3 x upper limit of normal (ULN) |
| ALT (SGPT) | ≥ 3 x ULN |
| Alkaline phosphatase | ≥ 3 x ULN |
| LDH | ≥ 3 x ULN |
| BUN | ≥ 30 mg/dL |
| Creatinine | ≥ 2.0 mg/dL |
| Uric Acid | |
| Men | $\geq 10.5 \text{ mg/dL}$ |
| Women | $\geq$ 8.5 mg/dL |
| Bilirubin (total) | $\geq 2.0 \text{ mg/dL}$ |
| CPK | ≥ 3 x ULN |
| Endocrinology | |
| Prolactin | > ULN |
| Hematology | |
| Hematocrit | |
| Men | $\leq$ 37 % and decrease of $\geq$ 3 percentage points from Baseline |
| Women | $\leq$ 32 % and decrease of $\geq$ 3 percentage points from Baseline |
| Hemoglobin | |
| Men | ≤ 11.5 g/dL |
| Women | ≤9.5 g/dL |
| White blood count | $\leq 2,800/ \text{ mm}^3 \text{ or } \geq 16,000/ \text{ mm}^3$ |
| Eosinophils | ≥ 10% |
| Neutrophils | ≤ 15% |
| Absolute neutrophil count | ≤ 1,000/ mm <sup>3</sup> |
| Platelet count $\leq 75,000/ \text{ mm}^3 \text{ or } \geq 700,000/ \text{ mm}^3$ | |
| Urinalysis | |
| Protein | Increase of $\geq 2$ units |
| Glucose | Increase of $\geq 2$ units |
| Additional Criteria | |
| Chloride | $\leq$ 90 mEq/L or $\geq$ 118 mEq/L |
| Potassium | $\leq 2.5 \text{ mEq/L or} \geq 6.5 \text{ mEq/L}$ |
| Sodium | $\leq 126 \text{ mEq/L or} \geq 156 \text{ mEq/L}$ |
| Calcium | $\leq$ 8.2 mg/dL or $\geq$ 12 mg/dL |
| Glucose | |
| Fasting | ≥ 100 mg/dL |
| Non-Fasting | ≥ 200 mg/dL |
| Total Cholesterol, Fasting ≥ 240 mg/dL | |
| LDL Cholesterol, Fasting ≥ 160 mg/dL | |
| HDL Cholesterol, Fasting | |
| Men | < 40 mg/dL |
| Women | < 50 mg/dL |
| Triglycerides, Fasting | $\geq 150 \text{ mg/dL}$ |
## Appendix 3 Criteria for Identifying ECG Measurements of Potential Clinical Relevance

| Variable | Criterion Value <sup>a</sup> | Change Relative to Baseline <sup>a</sup> |
|---|---|---|
| Heart Rate | ≥ 120 bpm | increase of $\geq 15$ bpm |
| | ≤ 50 bpm | decrease of $\geq$ 15 bpm |
| PR | ≥ 200 msec | increase of $\geq 50$ msec |
| QRS | ≥ 120 msec | increase of ≥ 20 msec |
| QTcF | > 450 msec | |
| | (males and females) | |

<sup>&</sup>lt;sup>a</sup>In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.

## **Appendix 4 Adverse Events of Interest**

| Appendix 4 Adverse Events of Interest | |
|---|---|
| AE Category | Preferred Term |
| EFFECT ON GLUCOSE | Blood glucose abnormal |
| | Blood glucose increased |
| | Diabetes mellitus |
| | Diabetes mellitus inadequate control |
| | Diabetes with hyperosmolarity |
| | Diabetic coma |
| | Diabetic hyperglycaemic coma |
| | Diabetic hyperosmolar coma |
| | Diabetic ketoacidosis |
| | Diabetic ketoacidotic hyperglycaemic coma |
| | Glucose tolerance decreased |
| | Glucose tolerance impaired |
| | Glucose tolerance test abnormal |
| | Glucose urine present |
| | Glycosuria |
| | Glycosylated haemoglobin increased |
| | Hyperglycaemia |
| | Hyperglycaemic hyperosmolar nonketotic syndrome |
| | Impaired fasting glucose |
| | Increased insulin requirement |
| | Indeterminate glucose tolerance |
| | Insulin resistance |
| | Insulin resistant diabetes |
| | Insulin tolerance test abnormal |
| | Insulin-requiring type 2 diabetes mellitus |
| | Ketoacidosis |
| | Ketonuria |
| | Ketosis |
| | Metabolic syndrome |
| | Type 1 diabetes mellitus |
| | Type 2 diabetes mellitus |
| | Urine ketone body present |
| EFFECT ON LIPIDS | 3-hydroxyacetyl-coenzyme A dehydrogenase deficiency |
| | Acquired mixed hyperlipidaemia |
| | Apolipoprotein |
| | Apolipoprotein A-I |
| | Apolipoprotein A-I abnormal |
| | Apolipoprotein A-I decreased |
| | Apolipoprotein A-I increased |
| | Apolipoprotein A-I normal |
| | Apolipoprotein A-II |
| | Apolipoprotein A-II abnormal |
| | Apolipoprotein A-II decreased |
| | Apolipoprotein A-II increased |
| | Apolipoprotein A-II normal |
| | A Time of D |

Statistical Analysis Plan 37 of 105 Version: 1.0 Date: 08/10/2022

Apolipoprotein B Apolipoprotein B abnormal Apolipoprotein B decreased Apolipoprotein B increased Apolipoprotein B normal

Apolipoprotein B/Apolipoprotein A-1 ratio

Apolipoprotein B/Apolipoprotein A-1 ratio increased

Apolipoprotein C

Apolipoprotein C abnormal

Apolipoprotein E

Apolipoprotein E abnormal

Apolipoprotein E increased

Apolipoprotein abnormal

Apolipoprotein decreased

Apolipoprotein increased

Apolipoprotein normal

Autoimmune hyperlipidaemia

Barth syndrome

Blood cholesterol

Blood cholesterol abnormal

Blood cholesterol decreased

Blood cholesterol esterase increased

Blood cholesterol increased

Blood cholesterol normal

Blood triglycerides

Blood triglycerides abnormal

Blood triglycerides decreased

Blood triglycerides increased

Blood triglycerides normal

Body fat disorder

CANDLE syndrome

Cardiac steatosis

Carnitine

Carnitine abnormal

Carnitine decreased

Carnitine deficiency

Carnitine increased

Carnitine normal

Carnitine palmitoyltransferase deficiency

Carnitine-acylcarnitine translocase deficiency

Cholesterol absorption efficiency decreased

Cholesterosis

Chylomicron decreased

Chylomicron increased

Chylomicrons

Congenital carnitine deficiency

Dyslipidaemia

Epidural lipomatosis

Facial wasting

Familial high density lipoprotein deficiency

Version: 1.0 Date: 08/10/2022

Familial hypertriglyceridaemia

Fat redistribution

Fatty acid deficiency

Fatty acid oxidation disorder

Fatty liver alcoholic

Free fatty acids

Free fatty acids abnormal

Free fatty acids decreased

Free fatty acids increased

Gastric xanthoma

HIV lipodystrophy

Hepatic steato-fibrosis

Hepatic steatosis

High density lipoprotein

High density lipoprotein abnormal

High density lipoprotein decreased

High density lipoprotein increased

High density lipoprotein normal

Hyper HDL cholesterolaemia

Hypercholesterolaemia

\*\*

Hyperchylomicronaemia

Hyperlipidaemia

Hypertriglyceridaemia

Hypo HDL cholesterolaemia

Hypocarnitinaemia

Hypocholesterolaemia

Hypolipidaemia

Hypotriglyceridaemia

Inborn error of lipid metabolism

Intermediate density lipoprotein decreased

Intermediate density lipoprotein increased

Intestinal lipomatosis

Intestinal steatosis

LDL/HDL ratio

LDL/HDL ratio decreased

LDL/HDL ratio increased

Lecithin-cholesterol acyltransferase activity decreased

Lecithin-cholesterol acyltransferase activity increased

Lecithin-cholesterol acyltransferase deficiency

Lipaemia retinalis

Lipaemic index score

Lipid metabolism disorder

Lipid proteinosis

Lipids

Lipids abnormal

Lipids decreased

Lipids increased

Lipids normal

Lipoatrophy

Lipodystrophy acquired

Lipoedema

Lipohypertrophy

Lipomatosis

Lipoprotein (a)

Lipoprotein (a) abnormal

Lipoprotein (a) decreased

Lipoprotein (a) increased

Lipoprotein (a) normal

Lipoprotein abnormal

Lipoprotein deficiency

Lipoprotein increased

Long-chain acyl-coenzyme A dehydrogenase deficiency

Low density lipoprotein

Low density lipoprotein abnormal

Low density lipoprotein decreased

Low density lipoprotein increased

Low density lipoprotein normal

Medium-chain acyl-coenzyme A dehydrogenase deficiency

Mesangiolipidosis

Non-alcoholic steatohepatitis

Non-high-density lipoprotein cholesterol

Non-high-density lipoprotein cholesterol decreased

Non-high-density lipoprotein cholesterol increased

Nonalcoholic fatty liver disease

Pancreatic steatosis

Parotid lipomatosis

Partial lipodystrophy

Phospholipidosis

Phytanic acid increased

Phytosterol level

Phytosterol level increased

Phytosterolaemia

Primary hypercholesterolaemia

Remnant hyperlipidaemia

Remnant-like lipoprotein particles

Remnant-like lipoprotein particles increased

Renal lipomatosis

Renal phospholipidosis

Serum pristanic acid increased

Short-chain acyl-coenzyme A dehydrogenase deficiency

Steatohepatitis

Tangier disease

Thyroid steatosis

Total cholesterol/HDL ratio

Total cholesterol/HDL ratio abnormal

Total cholesterol/HDL ratio decreased

Total cholesterol/HDL ratio increased

Total cholesterol/HDL ratio normal

Trifunctional protein deficiency

Type I hyperlipidaemia

Type II hyperlipidaemia

Type III hyperlipidaemia

Type IIa hyperlipidaemia

Type IIb hyperlipidaemia

Type IV hyperlipidaemia

Type V hyperlipidaemia

Very long-chain acyl-coenzyme A dehydrogenase deficiency


Very low density lipoprotein

Very low density lipoprotein abnormal

Very low density lipoprotein decreased

Very low density lipoprotein increased

Very low density lipoprotein normal

Xanthelasma

Xanthoma

Xanthomatosis

Zieve syndrome

EFFECTS ON WEIGHT

**EPS** 

Abnormal weight gain Body mass index abnormal Body mass index increased

Obesity

Overweight

Waist circumference increased

Weight fluctuation

Weight increased

Abnormal involuntary movement scale

Action tremor
Akathisia
Akinesia
Asterixis
Athetosis
Ballismus
Blepharospasm
Bradykinesia
Bradyphrenia

Buccoglossal syndrome

Chorea

Choreoathetosis Chronic tic disorder

Clumsiness Cogwheel rigidity Complex tic

Dopamine dysregulation syndrome

Drooling Dysarthria Dyskinesia

Dyskinesia neonatal Dyskinesia oesophageal

Dyslalia
Dysphonia
Dystonia
Dystonic tremor
Emprosthotonus
Essential tremor
Excessive eye blinking
Extrapyramidal disorder

Facial spasm

Fine motor skill dysfunction Freezing phenomenon

Fumbling
Gait disturbance
Gait inability
Gaze palsy

Glabellar reflex abnormal

Grimacing Head titubation Huntington's disease

Hyperkinesia

Hyperkinesia neonatal

Hypertonia

Hypertonia neonatal

Hypokinesia

Hypokinesia neonatal

Hypokinetic dysarthria

Intention tremor

Laryngeal tremor

Laryngospasm

Meige's syndrome

Micrographia

Mobility decreased

Motor dysfunction

Movement disorder

Muscle contractions involuntary

Muscle contracture

Muscle rigidity

Muscle spasms

Muscle spasticity

Muscle tightness

Muscle tone disorder

Muscle twitching

Musculoskeletal stiffness

Myoclonus

Myotonia

Nuchal rigidity

Oculogyric crisis

Oesophageal spasm

On and off phenomenon

Opisthotonus

Oromandibular dystonia

Oropharyngeal spasm

Parkinson's disease

Parkinson's disease psychosis

Parkinsonian crisis

Parkinsonian gait

Parkinsonian rest tremor

Parkinsonism

Parkinsonism hyperpyrexia syndrome

Periodic limb movement disorder

Pharyngeal dyskinesia

Pharyngeal dystonia

Pleurothotonus

Postural reflex impairment

Postural tremor

Posture abnormal

Posturing

Propulsive gait

Protrusion tongue

Provisional tic disorder

Psychomotor hyperactivity


Rabbit syndrome

Reduced facial expression

Respiratory dyskinesia

Resting tremor

Restless legs syndrome

Restlessness

Risus sardonicus

Saliva altered

Salivary hypersecretion

Secondary tic

Spasmodic dysphonia

Tardive dyskinesia

Tic

Tongue paralysis

Tongue spasm

Torticollis

Torticollis psychogenic

Tremor

Tremor neonatal

Trismus

Uvular spasm

Walking disability

Writer's cramp

5q minus syndrome

ABO haemolytic disease of newborn

ABO incompatibility

ADAMTS13 activity abnormal

ADAMTS13 activity assay

ADAMTS13 activity decreased

ADAMTS13 activity increased

ADAMTS13 activity normal

ADAMTS13 inhibitor screen assay

Aase syndrome

Abdominal lymphadenopathy

Abnormal clotting factor

Accessory spleen

Acid haemolysin test

Acid haemolysin test negative

Acid haemolysin test positive

Acquired Von Willebrand's disease

Acquired amegakaryocytic thrombocytopenia

Acquired antithrombin III deficiency

Acquired asplenia

Acquired complement deficiency disease

Acquired dysfibrinogenaemia

Acquired factor IX deficiency

Acquired factor VIII deficiency

Acquired factor XI deficiency

Acquired haemoglobinopathy

Acquired haemophilia

Acquired protein S deficiency

Acquired thalassaemia

Acral angiokeratoma-like pseudolymphoma


Activated partial thromboplastin time

HAEMATOPOIETIC/LEUKOPENIA

Activated partial thromboplastin time abnormal

Activated partial thromboplastin time normal

Activated partial thromboplastin time prolonged

Activated partial thromboplastin time ratio

Activated partial thromboplastin time ratio abnormal

Activated partial thromboplastin time ratio decreased

Activated partial thromboplastin time ratio fluctuation

Activated partial thromboplastin time ratio increased

Activated partial thromboplastin time ratio normal

Activated partial thromboplastin time shortened

Activated protein C resistance

Activated protein C resistance test

Activated protein C resistance test positive

Acute bilineal leukaemia

Acute biphenotypic leukaemia

Acute chest syndrome

Acute erythroid leukaemia

Acute febrile neutrophilic dermatosis

Acute haemolytic transfusion reaction

Acute haemorrhagic oedema of infancy

Acute leukaemia

Acute leukaemia in remission

Acute lymphocytic leukaemia

Acute lymphocytic leukaemia (in remission)

Acute lymphocytic leukaemia recurrent

Acute lymphocytic leukaemia refractory

Acute megakaryocytic leukaemia

Acute megakaryocytic leukaemia (in remission)

Acute monocytic leukaemia

Acute monocytic leukaemia (in remission)

Acute myeloid leukaemia

Acute myeloid leukaemia (in remission)

Acute myeloid leukaemia recurrent

Acute myeloid leukaemia refractory

Acute myelomonocytic leukaemia Acute promyelocytic leukaemia

Acute undifferentiated leukaemia

Adenoiditis

Administration site lymphadenopathy

Adult T-cell lymphoma/leukaemia

Adult T-cell lymphoma/leukaemia recurrent

Adult T-cell lymphoma/leukaemia refractory

Adult T-cell lymphoma/leukaemia stage I

Adult T-cell lymphoma/leukaemia stage II

Adult T-cell lymphoma/leukaemia stage III

Adult T-cell lymphoma/leukaemia stage IV

Agranulocytosis

Aleukaemic leukaemia

Allergic bronchopulmonary mycosis

Allergic eosinophilia

Alloimmunisation

Alpha-thalassaemia-intellectual deficit syndrome


Amegakaryocytic thrombocytopenia

Anaemia

Anaemia Heinz body

Anaemia folate deficiency

Anaemia macrocytic

Anaemia megaloblastic

Anaemia neonatal

Anaemia of chronic disease

Anaemia of malignant disease

Anaemia of pregnancy

Anaemia postoperative

Anaemia splenic

Anaemia vitamin B12 deficiency

Anaemia vitamin B6 deficiency

Anaemic hypoxia

Anaphylactoid syndrome of pregnancy

Anaplastic large cell lymphoma T- and null-cell types

Anaplastic large cell lymphoma T- and null-cell types recurrent

Anaplastic large cell lymphoma T- and null-cell types refractory

Anaplastic large cell lymphoma T- and null-cell types stage I

Anaplastic large cell lymphoma T- and null-cell types stage II

Anaplastic large cell lymphoma T- and null-cell types stage III

Anaplastic large cell lymphoma T- and null-cell types stage IV

Anaplastic large-cell lymphoma

Angiocentric lymphoma

Angiocentric lymphoma recurrent

Angiocentric lymphoma refractory

Angiocentric lymphoma stage I

Angiocentric lymphoma stage II

Angiocentric lymphoma stage III

Angiocentric lymphoma stage IV

Angioimmunoblastic T-cell lymphoma

Angioimmunoblastic T-cell lymphoma recurrent

Angioimmunoblastic T-cell lymphoma refractory

Angioimmunoblastic T-cell lymphoma stage I

Angioimmunoblastic T-cell lymphoma stage II Angioimmunoblastic T-cell lymphoma stage III

Angioimmunoblastic T-cell lymphoma stage IV

Angiolymphoid hyperplasia with eosinophilia

Anisochromia

Anisocytosis

Anti A antibody

Anti A antibody positive

Anti B antibody

Anti B antibody positive

Anti Kell antibody test

Anti Kell antibody test negative

Anti Kell antibody test positive

Anti factor IX antibody

Anti factor IX antibody increased

Anti factor IX antibody negative

Anti factor IX antibody positive

Anti factor V antibody

Anti factor V antibody positive

Anti factor VII antibody positive

Anti factor VIII antibody increased

Anti factor VIII antibody negative

Anti factor VIII antibody positive

Anti factor VIII antibody test

Anti factor X activity

Anti factor X activity abnormal

Anti factor X activity decreased

Anti factor X activity increased

Anti factor X activity normal

Anti factor X antibody

Anti factor X antibody negative

Anti factor X antibody positive

Anti factor XI antibody positive

Anti factor XII antibody positive

Anti factor Xa activity decreased

Anti factor Xa assay normal

Anti-complement antibody

Anti-erythropoietin antibody

Anti-erythropoietin antibody negative

Anti-erythropoietin antibody positive

Anti-prothrombin antibody positive

Anti-thrombin antibody

Antiphospholipid syndrome

Antithrombin III

Antithrombin III abnormal

Antithrombin III decreased

Antithrombin III deficiency

Antithrombin III increased

Aplasia pure red cell

Aplastic anaemia

Application site lymphadenopathy

Aspiration bone marrow

Aspiration bone marrow abnormal

Aspiration bone marrow normal

Asplenia

Atypical haemolytic uraemic syndrome

Atypical lymphocytic lobular panniculitis

Atypical mycobacterial lymphadenitis

Autoimmune anaemia

Autoimmune aplastic anaemia

Autoimmune haemolytic anaemia

Autoimmune heparin-induced thrombocytopenia

Autoimmune lymphoproliferative syndrome

Autoimmune neutropenia

Autoimmune pancytopenia

Autosomal recessive megaloblastic anaemia


Axillary web syndrome

B precursor type acute leukaemia

B-cell aplasia

B-cell lymphoma

B-cell lymphoma recurrent

B-cell lymphoma refractory

B-cell lymphoma stage I

B-cell lymphoma stage II

B-cell lymphoma stage III

B-cell lymphoma stage IV

B-cell prolymphocytic leukaemia

B-cell small lymphocytic lymphoma

B-cell small lymphocytic lymphoma recurrent

B-cell small lymphocytic lymphoma refractory

B-cell small lymphocytic lymphoma stage I

B-cell small lymphocytic lymphoma stage II

B-cell small lymphocytic lymphoma stage III

B-cell small lymphocytic lymphoma stage IV

B-cell type acute leukaemia

B-cell unclassifiable lymphoma high grade

B-cell unclassifiable lymphoma low grade

B-lymphocyte abnormalities

B-lymphocyte count

B-lymphocyte count abnormal

B-lymphocyte count decreased

B-lymphocyte count increased

Babesiosis

Band neutrophil count

Band neutrophil count decreased

Band neutrophil count increased

Band neutrophil percentage

Band neutrophil percentage decreased

Band neutrophil percentage increased

Bandaemia

Banti's syndrome

Basophil count

Basophil count abnormal

Basophil count decreased

Basophil count increased

Basophil count normal

Basophil morphology

Basophil morphology abnormal

Basophil morphology normal

Basophil percentage

Basophil percentage decreased

Basophil percentage increased

Basophilia

Basophilopenia

Benign ethnic neutropenia

Benign lymph node neoplasm

Benign neoplasm of thymus

Benign spleen tumour

Benjamin syndrome

Bernard-Soulier syndrome

Beta globin abnormal

Bicytopenia

Bing-Neel syndrome

Biopsy bone marrow

Biopsy bone marrow abnormal

Biopsy bone marrow normal

Biopsy lymph gland

Biopsy lymph gland abnormal

Biopsy lymph gland normal

Biopsy spleen

Biopsy spleen abnormal

Biopsy spleen normal

Biopsy thymus gland

Biopsy thymus gland abnormal

Biopsy thymus gland normal

Blackwater fever

Blast cell count decreased

Blast cell count increased

Blast cell crisis

Blast cell proliferation

Blast cells

Blast cells absent

Blast cells present

Blast crisis in myelogenous leukaemia

Blastic plasmacytoid dendritic cell neoplasia

Bleeding time

Bleeding time abnormal

Bleeding time normal

Bleeding time prolonged

Bleeding time shortened

Blood count

Blood count abnormal

Blood count normal

Blood disorder

Blood erythropoietin

Blood erythropoietin abnormal

Blood erythropoietin decreased

Blood erythropoietin increased

Blood erythropoietin normal

Blood fibrinogen

Blood fibrinogen abnormal

Blood fibrinogen decreased

Blood fibrinogen increased

Blood fibrinogen normal

Blood group A

Blood group AB

Blood group B

Blood group O

Blood grouping

Blood incompatibility haemolytic anaemia of newborn


Blood loss anaemia

Blood loss anaemia neonatal

Blood loss assessment

Blood thrombin

Blood thrombin abnormal

Blood thrombin decreased

Blood thrombin increased

Blood thrombin normal

Blood thromboplastin

Blood thromboplastin abnormal

Blood thromboplastin decreased

Blood thromboplastin increased

Blood thromboplastin normal

Blood type incompatibility

Blood viscosity abnormal

Blood viscosity decreased

Blood viscosity increased

Bone marrow band neutrophil count increased

Bone marrow basophilic leukocyte count increased

Bone marrow disorder

Bone marrow eosinophilic leukocyte count increased

Bone marrow failure

Bone marrow granuloma

Bone marrow haemorrhage

Bone marrow infiltration

Bone marrow ischaemia

Bone marrow leukaemic cell infiltration

Bone marrow metamyelocyte count increased

Bone marrow myelogram

Bone marrow myelogram abnormal

Bone marrow myelogram normal

Bone marrow necrosis

Bone marrow oedema

Bone marrow oedema syndrome

Bone marrow plasmacyte count increased

Bone marrow polymorphonuclear leukocyte count increased

Bone marrow reticulin fibrosis

Bone marrow transplant rejection

Bone marrow tumour cell infiltration

Breakthrough haemolysis

Breast implant-associated anaplastic large cell lymphoma

Broncholithiasis

Bronchopulmonary aspergillosis allergic

Burkitt's leukaemia

Burkitt's lymphoma

Burkitt's lymphoma recurrent

Burkitt's lymphoma refractory

Burkitt's lymphoma stage I

Burkitt's lymphoma stage II

Burkitt's lymphoma stage III

Burkitt's lymphoma stage IV

CANDLE syndrome

CD4 lymphocyte percentage decreased

CD4 lymphocyte percentage increased


CD4 lymphocytes

CD4 lymphocytes abnormal

CD4 lymphocytes decreased

CD4 lymphocytes increased

CD4 lymphocytes normal

CD4/CD8 ratio

CD4/CD8 ratio decreased

CD4/CD8 ratio increased

CD8 lymphocyte percentage decreased

CD8 lymphocyte percentage increased

CD8 lymphocytes

CD8 lymphocytes abnormal

CD8 lymphocytes decreased

CD8 lymphocytes increased

Capillary fragility abnormal

Capillary fragility decreased

Capillary fragility increased

Capillary fragility normal

Capillary fragility test

Capillary permeability

Capillary permeability increased

Capillary permeability normal

Carboxyhaemoglobinaemia

Cardiac haemolytic anaemia

Cardiac lymphangioma

Castleman's disease

Central nervous system leukaemia

Central nervous system lymphoma

Chediak-Higashi syndrome

Chloroma

Chloroma (in remission)

Chorea-acanthocytosis

Chronic eosinophilic leukaemia

Chronic granulomatous disease

Chronic leukaemia

Chronic leukaemia in remission

Chronic lymphocytic leukaemia

Chronic lymphocytic leukaemia (in remission)

Chronic lymphocytic leukaemia recurrent

Chronic lymphocytic leukaemia refractory

Chronic lymphocytic leukaemia stage 0

Chronic lymphocytic leukaemia stage 1 Chronic lymphocytic leukaemia stage 2

Chronic lymphocytic leukaemia stage 3

Chronic lymphocytic leukaemia stage 4

Chronic lymphocytic leukaemia transformation

Chronic myeloid leukaemia

Chronic myeloid leukaemia (in remission)

Chronic myeloid leukaemia recurrent

Chronic myeloid leukaemia transformation

Chronic myelomonocytic leukaemia

Chronic myelomonocytic leukaemia (in remission)

Chronic myelomonocytic leukaemia with N-ras gene mutation


Chronic pigmented purpura

Circulating anticoagulant

Circulating anticoagulant positive

Clonal haematopoiesis

Clot retraction

Clot retraction abnormal

Clot retraction normal

Clot retraction time prolonged

Clot retraction time shortened

Coagulation disorder neonatal

Coagulation factor

Coagulation factor IX level

Coagulation factor IX level abnormal

Coagulation factor IX level decreased

Coagulation factor IX level increased

Coagulation factor IX level normal

Coagulation factor V level

Coagulation factor V level abnormal

Coagulation factor V level decreased

Coagulation factor V level increased

Coagulation factor V level normal

Coagulation factor VII level

Coagulation factor VII level abnormal

Coagulation factor VII level decreased

Coagulation factor VII level increased

Coagulation factor VII level normal

Coagulation factor VIII level

Coagulation factor VIII level abnormal

Coagulation factor VIII level decreased

Coagulation factor VIII level increased

Coagulation factor VIII level normal

Coagulation factor X level

Coagulation factor X level abnormal

Coagulation factor X level decreased

Coagulation factor X level increased

Coagulation factor X level normal

Coagulation factor XI level

Coagulation factor XI level abnormal

Coagulation factor XI level decreased

Coagulation factor XI level increased

Coagulation factor XI level normal

Coagulation factor XII level

Coagulation factor XII level abnormal

Coagulation factor XII level decreased

Coagulation factor XII level increased

Coagulation factor XII level normal

Coagulation factor XIII level

Coagulation factor XIII level abnormal

Coagulation factor XIII level decreased

Coagulation factor XIII level increased

Coagulation factor XIII level normal

Coagulation factor decreased

Coagulation factor deficiency

Coagulation factor increased

Coagulation factor inhibitor assay

Coagulation factor level normal


Coagulation factor mutation

Coagulation test

Coagulation test abnormal

Coagulation test normal

Coagulation time

Coagulation time abnormal

Coagulation time normal

Coagulation time prolonged

Coagulation time shortened

Coagulopathy

Cold type haemolytic anaemia

Complement deficiency disease

Composite lymphoma

Congenital anaemia

Congenital aplastic anaemia

Congenital coagulopathy

Congenital dyserythropoietic anaemia

Congenital dysfibrinogenaemia

Congenital dyskeratosis

Congenital haematological disorder

Congenital hypercoagulation

Congenital hypotransferrinaemia

Congenital lymphatic dysplasia

Congenital lymphoedema

Congenital malaria

Congenital methaemoglobinaemia

Congenital thrombocyte disorder

Congenital thrombocytopenia

Congenital thymus absence

Congenital white blood cell disorder

Conjunctival lymphangiectasia

Conjunctival pallor

Coombs direct test

Coombs direct test negative

Coombs direct test positive

Coombs indirect test

Coombs indirect test negative

Coombs indirect test positive

Coombs negative haemolytic anaemia

Coombs positive haemolytic anaemia

Coombs test

Coombs test negative

Coombs test positive

Crossmatch

Crossmatch compatible

Crossmatch incompatible

Cutaneous B-cell lymphoma

Cutaneous T-cell dyscrasia

Cutaneous T-cell lymphoma

Cutaneous T-cell lymphoma recurrent

Cutaneous T-cell lymphoma refractory

Cutaneous T-cell lymphoma stage I

Cutaneous T-cell lymphoma stage II

Cutaneous T-cell lymphoma stage III

Cutaneous T-cell lymphoma stage IV

Cutaneous extramedullary haemopoiesis


Cutaneous lymphoma

Cutaneovisceral angiomatosis with thrombocytopenia

Cyclic neutropenia

Cystic lymphangioma

Cytomegalovirus mononucleosis

Cytopenia

Cytophagic histiocytic panniculitis

Deficiency anaemia

Delayed haematopoietic reconstitution

Delayed haemolytic transfusion reaction

Delayed serologic transfusion reaction

Delta-beta thalassaemia

Dermatopathic lymphadenopathy

Differential white blood cell count

Differential white blood cell count abnormal

Differential white blood cell count normal

Diffuse large B-cell lymphoma

Diffuse large B-cell lymphoma recurrent

Diffuse large B-cell lymphoma refractory

Diffuse large B-cell lymphoma stage I

Diffuse large B-cell lymphoma stage II

Diffuse large B-cell lymphoma stage III

Diffuse large B-cell lymphoma stage IV

Dilutional coagulopathy

Disseminated intravascular coagulation

Disseminated intravascular coagulation in newborn

Disseminated large cell lymphoma

Double heterozygous sickling disorders

Double hit lymphoma

Dubowitz syndrome

Dysglobulinaemia

Ecchymosis

Elephantiasis

Elephantiasis nostras verrucosa

Elliptocytosis

Elliptocytosis hereditary

Endothelial protein C receptor polymorphism

Engraftment syndrome

Enteritis leukopenic

Enteropathy-associated T-cell lymphoma

Eosinopenia

Eosinophil count

Eosinophil count abnormal

Eosinophil count decreased

Eosinophil count increased

Eosinophil count normal

Eosinophil morphology

Eosinophil morphology abnormal

Eosinophil morphology normal

Eosinophil percentage

Eosinophil percentage abnormal

Eosinophil percentage decreased

Eosinophil percentage increased


Eosinophilia

Eosinophilia myalgia syndrome

Eosinophilic bronchitis

Eosinophilic cellulitis

Eosinophilic colitis

Eosinophilic cystitis

Eosinophilic fasciitis

Eosinophilic gastritis

Eosinophilic granulomatosis with polyangiitis

Eosinophilic leukaemia

Eosinophilic myocarditis

Eosinophilic oesophagitis

Eosinophilic otitis media

Eosinophilic panniculitis

Eosinophilic pleural effusion

Eosinophilic pneumonia

Eosinophilic pneumonia acute

Eosinophilic pneumonia chronic

Eosinophilic pustular folliculitis

Eosinophilic pustulosis

Eosinophilic rhinitis

Epstein Barr virus positive mucocutaneous ulcer

Epstein-Barr virus associated lymphoma

Epstein-Barr virus associated lymphoproliferative disorder

Erdheim-Chester disease

Erythraemic myelosis (in remission)

Erythroblast count

Erythroblast count abnormal

Erythroblast count decreased

Erythroblast count increased

Erythroblast count normal

Erythroblast morphology

Erythroblast morphology abnormal

Erythroblastosis

Erythroblastosis foetalis

Erythrocyte osmotic fragility test

Erythroid maturation arrest

Erythroid series abnormal

Erythropenia

Erythrophagocytosis

Erythropoiesis abnormal

Erythropoietin deficiency anaemia

Erythrosis

Essential thrombocythaemia

Ethanol gelation test

Ethanol gelation test negative

Ethanol gelation test positive

Evans syndrome

Extramedullary haemopoiesis

Extranodal marginal zone B-cell lymphoma (BALT type)

Extranodal marginal zone B-cell lymphoma (MALT type)

Extranodal marginal zone B-cell lymphoma (MALT type) recurrent

Extranodal marginal zone B-cell lymphoma (MALT type) refractory


Extranodal marginal zone B-cell lymphoma (MALT type) stage I

Extranodal marginal zone B-cell lymphoma (MALT type) stage II

Extranodal marginal zone B-cell lymphoma (MALT type) stage III

Extranodal marginal zone B-cell lymphoma (MALT type) stage IV

Extravascular haemolysis

Factor I deficiency

Factor II deficiency

Factor II inhibition

Factor II mutation

Factor III deficiency

Factor IX deficiency

Factor IX inhibition

Factor V Leiden mutation

Factor V deficiency

Factor V inhibition

Factor VII deficiency

Factor VII inhibition

Factor VIII deficiency

Factor VIII inhibition

Factor X deficiency

Factor X inhibition

Factor XI deficiency

Factor XII deficiency

Factor XIII Inhibition

Factor XIII deficiency

Factor Xa activity abnormal

Factor Xa activity decreased

Factor Xa activity increased

Factor Xa activity normal

Factor Xa activity test

Familial haemophagocytic lymphohistiocytosis

Familial polycythaemia

Febrile bone marrow aplasia

Febrile neutropenia

Felty's syndrome

Fibrin

Fibrin D dimer

Fibrin D dimer decreased

Fibrin D dimer increased

Fibrin D dimer normal

Fibrin abnormal

Fibrin decreased

Fibrin degradation products

Fibrin degradation products increased

Fibrin degradation products normal

Fibrin increased

Fibrin normal

Fibrinogen degradation products increased


Fibrinolysis

Fibrinolysis abnormal

Fibrinolysis decreased

Fibrinolysis increased

Fibrinolysis normal

Filariasis lymphatic

Foetal anaemia

Foetal haemoglobin

Foetal haemoglobin decreased

Foetal haemoglobin increased

Foetal haemoglobin normal

Follicle centre lymphoma diffuse small cell lymphoma

Follicle centre lymphoma diffuse small cell lymphoma recurrent

Follicle centre lymphoma diffuse small cell lymphoma refractory

Follicle centre lymphoma diffuse small cell lymphoma stage I

Follicle centre lymphoma diffuse small cell lymphoma stage II

Follicle centre lymphoma diffuse small cell lymphoma stage III

Follicle centre lymphoma diffuse small cell lymphoma stage IV

Follicle centre lymphoma, follicular grade I, II, III

Follicle centre lymphoma, follicular grade I, II, III recurrent

Follicle centre lymphoma, follicular grade I, II, III refractory

Follicle centre lymphoma, follicular grade I, II, III stage I

Follicle centre lymphoma, follicular grade I, II, III stage II

Follicle centre lymphoma, follicular grade I, II, III stage III

Follicle centre lymphoma, follicular grade I, II, III stage IV

Follicular dendritic cell sarcoma

Follicular lymphoma

Follicular lymphoma stage I

Follicular lymphoma stage II

Follicular lymphoma stage III

Follicular lymphoma stage IV

Free haemoglobin

Free haemoglobin absent

Free haemoglobin present

Full blood count

Full blood count abnormal

Full blood count decreased

Full blood count increased

Full blood count normal

Gammopathy

Gastroenteritis eosinophilic

Gastrointestinal lymphoma

Gastrosplenic fistula

Gelatinous transformation of the bone marrow

Glanzmann's disease

Gleich's syndrome

Glucose-6-phosphate dehydrogenase

Glucose-6-phosphate dehydrogenase abnormal

Glucose-6-phosphate dehydrogenase deficiency


Glucose-6-phosphate dehydrogenase normal

Glutathione decreased

Glutathione increased

Glutathione synthetase deficiency

Glutathione test

Good syndrome

Granulocyte count

Granulocyte count decreased

Granulocyte count increased

Granulocyte percentage

Granulocytes abnormal

Granulocytes maturation arrest

Granulocytopenia

Granulocytopenia neonatal

Granulocytosis

Granulomatous T-cell pseudolymphoma

Granulomatous lymphadenitis

Grey zone lymphoma

HELLP syndrome

Haemangioma of spleen

Haemangioma-thrombocytopenia syndrome

Haematocrit

Haematocrit abnormal

Haematocrit decreased

Haematocrit increased

Haematocrit normal

Haematological malignancy

Haematology test

Haematology test abnormal

Haematology test normal

Haematopoietic neoplasm

Haematotoxicity

Haemoconcentration

Haemodilution

Haemoglobin

Haemoglobin A absent

Haemoglobin A present

Haemoglobin A2

Haemoglobin Barts absent

Haemoglobin Barts present

Haemoglobin C

Haemoglobin C disease

Haemoglobin C present

Haemoglobin C trait

Haemoglobin D disease

Haemoglobin D trait

Haemoglobin E

Haemoglobin E absent

Haemoglobin E disease

Haemoglobin E present

Haemoglobin E trait

Haemoglobin E-thalassaemia disease

Haemoglobin Lepore trait

Haemoglobin S

Haemoglobin S decreased

Haemoglobin S increased

Haemoglobin S normal

Haemoglobin abnormal

Haemoglobin decreased

Haemoglobin distribution width

Haemoglobin distribution width decreased

Haemoglobin distribution width increased


Haemoglobin electrophoresis

Haemoglobin electrophoresis abnormal

Haemoglobin electrophoresis normal

Haemoglobin increased

Haemoglobin normal

Haemoglobinaemia

Haemoglobinopathy

Haemoglobinuria

Haemolysis

Haemolysis neonatal

Haemolytic anaemia

Haemolytic anaemia enzyme specific

Haemolytic icteroanaemia

Haemolytic transfusion reaction

Haemolytic uraemic syndrome

Haemophagocytic lymphohistiocytosis

Haemophilia

Haemophilia A with anti factor VIII

Haemophilia A without inhibitors

Haemophilia B with anti factor IX

Haemophilia B without inhibitors

Haemophilic pseudotumour

Haemorrhagic diathesis

Haemorrhagic disease of newborn

Haemorrhagic disorder

Haemorrhagic vasculitis

Haemosiderinuria

Hairy cell leukaemia

Hairy cell leukaemia recurrent

Hand and foot syndrome secondary to sickle cell anaemia

Heavy chain disease

Heinz bodies

Henoch-Schonlein purpura

Henoch-Schonlein purpura nephritis

Heparin resistance

Heparin-induced thrombocytopenia

Heparin-induced thrombocytopenia test

Heparin-induced thrombocytopenia test positive

Hepatic infiltration eosinophilic

Hepatic lymphocytic infiltration

Hepatosplenic T-cell lymphoma

Hepatosplenic abscess

Hepatosplenic candidiasis

Hepatosplenomegaly

Hepatosplenomegaly neonatal

Hereditary haemolytic anaemia

Hereditary sideroblastic anaemia

Hereditary spherocytosis

Hereditary stomatocytosis

Hermansky-Pudlak syndrome

Hexokinase deficiency anaemia

High grade B-cell lymphoma Burkitt-like lymphoma

High grade B-cell lymphoma Burkitt-like lymphoma recurrent

High grade B-cell lymphoma Burkitt-like lymphoma refractory

High grade B-cell lymphoma Burkitt-like lymphoma stage I High grade B-cell lymphoma Burkitt-like lymphoma stage II High grade B-cell lymphoma Burkitt-like lymphoma stage III High grade B-cell lymphoma Burkitt-like lymphoma stage IV High-grade B-cell lymphoma

Hilar lymphadenopathy

Histiocytic medullary reticulosis

Histiocytic necrotising lymphadenitis

Histiocytic sarcoma

Histiocytosis

Hodgkin's disease

Hodgkin's disease lymphocyte depletion stage I site unspecified Hodgkin's disease lymphocyte depletion stage I subdiaphragm Hodgkin's disease lymphocyte depletion stage I supradiaphragm Hodgkin's disease lymphocyte depletion stage II site unspecified Hodgkin's disease lymphocyte depletion stage II subdiaphragm Hodgkin's disease lymphocyte depletion stage II supradiaphragm Hodgkin's disease lymphocyte depletion type recurrent Hodgkin's disease lymphocyte depletion type refractory Hodgkin's disease lymphocyte depletion type stage III Hodgkin's disease lymphocyte depletion type stage IV

Hodgkin's disease lymphocyte depletion type stage unspecified

Hodgkin's disease lymphocyte predominance stage I site unspec

Hodgkin's disease lymphocyte predominance stage I subdiaphragm

Hodgkin's disease lymphocyte predominance stage I supradiaphragm

Hodgkin's disease lymphocyte predominance stage II site unspec Hodgkin's disease lymphocyte predominance stage II subdiaphragm

Hodgkin's disease lymphocyte predominance stage II supradiaphragm

Hodgkin's disease lymphocyte predominance type recurrent

Hodgkin's disease lymphocyte predominance type refractory

Hodgkin's disease lymphocyte predominance type stage III

Hodgkin's disease lymphocyte predominance type stage IV

Hodgkin's disease lymphocyte predominance type stage unspecified

Hodgkin's disease mixed cellularity recurrent

Hodgkin's disease mixed cellularity refractory

Hodgkin's disease mixed cellularity stage I site unspecified

Hodgkin's disease mixed cellularity stage I subdiaphragmatic

Hodgkin's disease mixed cellularity stage I supradiaphragmatic

Hodgkin's disease mixed cellularity stage II subdiaphragmatic

Hodgkin's disease mixed cellularity stage II supradiaphragmatic


Hodgkin's disease mixed cellularity stage III

Hodgkin's disease mixed cellularity stage IV

Hodgkin's disease mixed cellularity stage unspecified

Hodgkin's disease nodular sclerosis

Hodgkin's disease nodular sclerosis recurrent

Hodgkin's disease nodular sclerosis refractory

Hodgkin's disease nodular sclerosis stage I

Hodgkin's disease nodular sclerosis stage II

Hodgkin's disease nodular sclerosis stage III

Hodgkin's disease nodular sclerosis stage IV

Hodgkin's disease recurrent

Hodgkin's disease refractory

Hodgkin's disease stage I

Hodgkin's disease stage II

Hodgkin's disease stage III

Hodgkin's disease stage IV

Hodgkin's disease unclassifiable

Hyperbilirubinaemia

Hyperchromasia

Hyperchromic anaemia

Hypercoagulation

Hypereosinophilic syndrome

Hyperfibrinogenaemia

Hyperfibrinolysis

Hypergammaglobulinaemia

Hypergammaglobulinaemia benign monoclonal

Hyperglobulinaemia

Hyperhomocysteinaemia

Hyperleukocytosis

Hyperplasia of thymic epithelium

Hyperprothrombinaemia

Hypersensitivity vasculitis

Hypersplenism

Hypersplenism congenital

Hyperthrombinaemia

Hyperviscosity syndrome

Hypochromasia

Hypochromic anaemia

Hypocoagulable state

Hypocomplementaemia

Hypofibrinogenaemia

Hypoglobulinaemia

Hypoplastic anaemia

Hypoprothrombinaemia

Hyposplenism

Hypothrombinaemia

Hypothromboplastinaemia

Hypotransferrinaemia

ISTH score for disseminated intravascular coagulation

Idiopathic CD4 lymphocytopenia

Idiopathic neutropenia

Immature granulocyte count

Immature granulocyte count increased

Immature granulocyte percentage increased

Immune thrombocytopenia

Immune-mediated cytopenia

Immunoblastic lymphoma

Increased tendency to bruise

Indeterminable ABO blood type

Infantile genetic agranulocytosis

Infantile scurvy

Infected lymphocele

Infectious mononucleosis

Infusion site lymphadenopathy

Injection site lymphadenopathy


International normalised ratio

International normalised ratio abnormal

International normalised ratio decreased

International normalised ratio fluctuation

International normalised ratio increased

International normalised ratio normal

Intestinal T-cell lymphoma recurrent

Intestinal T-cell lymphoma refractory

Intestinal T-cell lymphoma stage I

Intestinal T-cell lymphoma stage II

Intestinal T-cell lymphoma stage III

Intestinal T-cell lymphoma stage IV

Intravascular haemolysis

Iron deficiency anaemia

Isoimmune haemolytic disease

Jaundice

Jaundice acholuric

Jaundice neonatal

Jessner's lymphocytic infiltration

Juvenile chronic myelomonocytic leukaemia

Kell blood group positive

Lactescent serum

Langerhans cell sarcoma

Langerhans' cell histiocytosis

Large granular lymphocytosis

Leptomeningeal myelomatosis

Leukaemia

Leukaemia basophilic

Leukaemia cutis

Leukaemia granulocytic

Leukaemia in remission

Leukaemia monocytic

Leukaemia recurrent

Leukaemic cardiac infiltration

Leukaemic infiltration

Leukaemic infiltration extramedullary

Leukaemic infiltration gingiva

Leukaemic infiltration hepatic

Leukaemic infiltration ovary

Leukaemic infiltration pulmonary

Leukaemic infiltration renal

Leukaemic lymphoma

Leukaemic retinopathy

Leukaemoid reaction

Leukocyte adhesion deficiency type I

Leukocyte vacuolisation

Leukocytosis

Leukoerythroblastic anaemia

Leukoerythroblastosis

Leukopenia

Leukopenia neonatal

Leukostasis syndrome

Light chain disease

Lineage switch leukaemia

Loeffler's syndrome

Loefgren syndrome

Loss of CAR T-cell persistence

Lupus anticoagulant hypoprothrombinaemia syndrome

Lymph gland infection

Lymph node abscess

Lymph node calcification

Lymph node fibrosis

Lymph node haemorrhage

Lymph node pain

Lymph node rupture

Lymph node tuberculosis

Lymph node ulcer

Lymph nodes scan abnormal

Lymph nodes scan normal

Lymphadenitis

Lymphadenitis bacterial

Lymphadenitis fungal

Lymphadenitis helminthic

Lymphadenitis viral

Lymphadenocyst

Lymphadenopathy

Lymphadenopathy mediastinal

Lymphangiectasia

Lymphangiectasia intestinal

Lymphangiectasia intestinal congenital

Lymphangioleiomyomatosis

Lymphangioma

Lymphangiopathy

Lymphangiosarcoma

Lymphangiosis carcinomatosa

Lymphangitis

Lymphatic disorder

Lymphatic duct injury

Lymphatic fistula

Lymphatic insufficiency

Lymphatic obstruction

Lymphatic sinus catarrh

Lymphatic system neoplasm

Lymphoblast count

Lymphoblast count increased

Lymphoblast morphology

Lymphoblast morphology abnormal

Lymphoblast morphology normal

Lymphoblastosis

Lymphocele

Lymphocyte count

Lymphocyte count abnormal

Lymphocyte count decreased

Lymphocyte count increased

Lymphocyte count normal

Lymphocyte morphology

Lymphocyte morphology abnormal

Lymphocyte morphology normal

Lymphocyte percentage

Lymphocyte percentage abnormal

Lymphocyte percentage decreased

Lymphocyte percentage increased

Lymphocyte stimulation test

Lymphocyte stimulation test negative

Lymphocyte stimulation test positive

Lymphocyte transformation test

Lymphocyte transformation test negative

Lymphocyte transformation test positive

Lymphocyte/monocyte ratio decreased

Lymphocytic infiltration

Lymphocytic leukaemia

Lymphocytic lymphoma

Lymphocytic oesophagitis

Lymphocytopenia neonatal

Lymphocytosis

Lymphoedema

Lymphogranuloma venereum

Lymphoid hyperplasia of intestine

Lymphoid leukaemia (in remission)

Lymphoid tissue hyperplasia

Lymphoid tissue hypoplasia

Lymphoma

Lymphoma AIDS related

Lymphoma transformation

Lymphopenia

Lymphoplasia

Lymphoplasmacytoid lymphoma/immunocytoma

Lymphoplasmacytoid lymphoma/immunocytoma recurrent

Lymphoplasmacytoid lymphoma/immunocytoma refractory

Lymphoplasmacytoid lymphoma/immunocytoma stage I

Lymphoplasmacytoid lymphoma/immunocytoma stage II

Lymphoplasmacytoid lymphoma/immunocytoma stage III Lymphoplasmacytoid lymphoma/immunocytoma stage IV

Lymphoproliferative disorder

Lymphoproliferative disorder in remission

Lymphorrhoea

Lymphostasis

MLASA syndrome

MNS system antibodies positive

MYH9-related disease

Macrocytosis

Macrophage count

Macrophages decreased

Macrophages increased

Malaria

Malaria recrudescence

Malaria relapse

Malignant histiocytosis

Malignant lymphoid neoplasm

Malignant lymphoma unclassifiable high grade

Malignant lymphoma unclassifiable low grade

Malignant mast cell neoplasm

Malignant neoplasm of thymus

Malignant splenic neoplasm

Mantle cell lymphoma

Mantle cell lymphoma recurrent

Mantle cell lymphoma refractory

Mantle cell lymphoma stage I

Mantle cell lymphoma stage II

Mantle cell lymphoma stage III

Mantle cell lymphoma stage IV

March haemoglobinuria

Marginal zone lymphoma

Marginal zone lymphoma recurrent

Marginal zone lymphoma refractory

Marginal zone lymphoma stage I

Marginal zone lymphoma stage II

Marginal zone lymphoma stage III

Marginal zone lymphoma stage IV

Marrow hyperplasia

Mast cell activation syndrome

Mastocytic leukaemia

Mastocytosis

Mature B-cell type acute leukaemia

McLeod neuroacanthocytosis syndrome

Mean cell haemoglobin

Mean cell haemoglobin concentration

Mean cell haemoglobin concentration abnormal

Mean cell haemoglobin concentration decreased

Mean cell haemoglobin concentration increased Mean cell haemoglobin concentration normal

Mean cell haemoglobin decreased

Mean cell haemoglobin increased

Mean cell haemoglobin normal

Mean cell volume

Mean cell volume abnormal

Mean cell volume decreased

Mean cell volume increased

Mean cell volume normal

Mean platelet volume

Mean platelet volume abnormal

Mean platelet volume decreased

Mean platelet volume increased

Mean platelet volume normal

Medical device site lymphadenopathy

Megakaryocyte destruction increased


Megakaryocytes

Megakaryocytes abnormal

Megakaryocytes decreased

Megakaryocytes increased

Megakaryocytes normal

Megaloblasts increased

Melanaemia

Meningitis eosinophilic

Metamyelocyte count

Metamyelocyte count decreased

Metamyelocyte count increased

Metamyelocyte percentage

Metamyelocyte percentage increased

Metastases to bone marrow

Metastases to lymph nodes

Metastases to spleen

Metastatic lymphoma

Methaemoglobinaemia

Methaemoglobinuria

Methylenetetrahydrofolate reductase deficiency

Methylenetetrahydrofolate reductase polymorphism

Microangiopathic haemolytic anaemia

Microcytic anaemia

Microcytosis

Minimal residual disease

Mitogen stimulation test

Mitogen stimulation test abnormal

Mitogen stimulation test normal

Monoblast count

Monoblast count decreased

Monoblast count increased

Monoclonal B-cell lymphocytosis

Monoclonal gammopathy

Monocyte count

Monocyte count abnormal

Monocyte count decreased

Monocyte count increased

Monocyte count normal

Monocyte morphology

Monocyte morphology abnormal

Monocyte percentage

Monocyte percentage abnormal

Monocyte percentage decreased

Monocyte percentage increased

Monocytic leukaemia in remission

Monocytopenia

Monocytosis

Mononuclear cell count

Mononuclear cell count abnormal

Mononuclear cell count decreased

Mononuclear cell count increased

Mononuclear cell percentage

Mononucleosis syndrome

Multicentric reticulohistiocytosis

Myeloblast count

Myeloblast count decreased

Myeloblast count increased

Myeloblast percentage

Myeloblast percentage decreased

Myeloblast percentage increased

Myeloblast present

Myeloblastoma

Myelocyte count

Myelocyte count decreased

Myelocyte count increased

Myelocyte percentage

Myelocyte percentage decreased

Myelocyte percentage increased

Myelocyte present

Myelocytosis

Myelodysplastic syndrome

Myelodysplastic syndrome transformation

Myelodysplastic syndrome unclassifiable

Myelofibrosis

Myeloid leukaemia

Myeloid leukaemia in remission

Myeloid maturation arrest

Myeloid metaplasia

Myelolipoma

Myeloperoxidase deficiency

Myeloproliferative neoplasm

Myelosuppression

Natural killer T cell count

Natural killer T cell count decreased

Natural killer T cell count increased

Natural killer cell count

Natural killer cell count decreased

Natural killer cell count increased

Natural killer-cell leukaemia

Natural killer-cell lymphoblastic lymphoma

Necrotic lymphadenopathy

Neonatal alloimmune thrombocytopenia

Neonatal leukaemia

Neoplasm of thymus

Nephrogenic anaemia

Neuroacanthocytosis

Neutropenia

Neutropenia neonatal

Neutropenic colitis

Neutropenic infection

Neutropenic sepsis

Neutrophil Fc gamma RIIIb deficiency

Neutrophil Pelger-Huet anomaly present

Neutrophil chemotaxis

Neutrophil chemotaxis abnormal

Neutrophil chemotaxis normal

Neutrophil count

Neutrophil count abnormal

Neutrophil count decreased

Neutrophil count increased

Neutrophil count normal

Neutrophil function disorder


Neutrophil function test

Neutrophil function test abnormal

Neutrophil function test normal

Neutrophil hypersegmented morphology present

Neutrophil morphology

Neutrophil morphology abnormal

Neutrophil morphology normal

Neutrophil percentage

Neutrophil percentage abnormal

Neutrophil percentage decreased

Neutrophil percentage increased

Neutrophil toxic granulation present

Neutrophil/lymphocyte ratio

Neutrophil/lymphocyte ratio decreased

Neutrophil/lymphocyte ratio increased

Neutrophilia

Neutrophilic dermatosis

Nodal marginal zone B-cell lymphoma

Nodal marginal zone B-cell lymphoma recurrent

Nodal marginal zone B-cell lymphoma refractory

Nodal marginal zone B-cell lymphoma stage I

Nodal marginal zone B-cell lymphoma stage II

Nodal marginal zone B-cell lymphoma stage III

Nodal marginal zone B-cell lymphoma stage IV

Nodular lymphocyte predominant Hodgkin lymphoma

Non-Hodgkin's lymphoma

Non-Hodgkin's lymphoma metastatic

Non-Hodgkin's lymphoma recurrent

Non-Hodgkin's lymphoma refractory

Non-Hodgkin's lymphoma stage I

Non-Hodgkin's lymphoma stage II

Non-Hodgkin's lymphoma stage III

Non-Hodgkin's lymphoma stage IV

Non-Hodgkin's lymphoma transformed recurrent

Non-Hodgkin's lymphoma unspecified histology aggressive

Non-Hodgkin's lymphoma unspecified histology aggressive recurrent

Non-Hodgkin's lymphoma unspecified histology aggressive refractory

Non-Hodgkin's lymphoma unspecified histology aggressive stage I

Non-Hodgkin's lymphoma unspecified histology aggressive stage II

Non-Hodgkin's lymphoma unspecified histology aggressive stage III

Non-Hodgkin's lymphoma unspecified histology aggressive stage IV

Non-Hodgkin's lymphoma unspecified histology indolent

Non-Hodgkin's lymphoma unspecified histology indolent stage I

Non-Hodgkin's lymphoma unspecified histology indolent stage II

Non-Hodgkin's lymphoma unspecified histology indolent stage III

Non-Hodgkin's lymphoma unspecified histology indolent stage IV


Non-immune heparin associated thrombocytopenia

Nontherapeutic agent blood negative

Nontherapeutic agent blood positive

Normochromic anaemia

Normochromic normocytic anaemia

Normocytic anaemia

Nucleated red cells

Ocular icterus

Ocular lymphoma

Oculoglandular syndrome

Omenn syndrome

Oral purpura

Oropharyngeal lymphoid hyperplasia

PFAPA syndrome

POEMS syndrome

PSTPIP1-associated myeloid-related proteinaemia inflammatory

syndrome

Pancytopenia

Panmyelopathy

Paraproteinaemia

Paratracheal lymphadenopathy

Paroxysmal nocturnal haemoglobinuria

Passenger lymphocyte syndrome

Pearson's syndrome

Peripheral T-cell lymphoma unspecified

Peripheral T-cell lymphoma unspecified recurrent

Peripheral T-cell lymphoma unspecified refractory

Peripheral T-cell lymphoma unspecified stage I

Peripheral T-cell lymphoma unspecified stage II

Peripheral T-cell lymphoma unspecified stage III

Peripheral T-cell lymphoma unspecified stage IV

Perisplenitis

Pernicious anaemia

Persistent generalised lymphadenopathy

Petechiae

Philadelphia positive acute lymphocytic leukaemia

Philadelphia positive chronic myeloid leukaemia

Pickwickian syndrome

Pigment nephropathy

Placental transfusion syndrome

Plasma cell count

Plasma cell disorder

Plasma cell leukaemia

Plasma cell leukaemia in remission

Plasma cell myeloma

Plasma cell myeloma in remission

Plasma cell myeloma recurrent

Plasma cell myeloma refractory

Plasma cells absent

Plasma cells decreased

Plasma cells increased

Plasma cells present

Plasma viscosity

Plasma viscosity abnormal

Plasma viscosity decreased

Plasma viscosity normal

Plasmablast count

Plasmablast count decreased

Plasmablast count increased


Plasmablastic lymphoma

Plasmacytoma

Plasmacytosis

Plasmin decreased

Plasmin increased

Plasmin inhibitor

Plasmin inhibitor decreased

Plasmin inhibitor increased

Plasminogen

Plasminogen activator inhibitor

Plasminogen activator inhibitor decreased

Plasminogen activator inhibitor increased

Plasminogen activator inhibitor polymorphism

Plasminogen activator inhibitor type 1 deficiency

Plasminogen decreased

Plasminogen increased

Plasminogen normal

Plasmodium falciparum infection

Plasmodium knowlesi infection

Plasmodium malariae infection

Plasmodium ovale infection

Plasmodium vivax infection

Platelet adhesiveness

Platelet adhesiveness abnormal

Platelet adhesiveness decreased

Platelet adhesiveness increased

Platelet adhesiveness normal

Platelet aggregation abnormal

Platelet aggregation decreased

Platelet aggregation increased

Platelet aggregation inhibition Platelet aggregation normal

Platelet aggregation test

Platelet anisocytosis

Platelet count

Platelet count abnormal

Platelet count decreased

Platelet count increased

Platelet count normal

Platelet destruction increased

Platelet disorder

Platelet distribution width

Platelet distribution width abnormal

Platelet distribution width decreased

Platelet distribution width increased

Platelet dysfunction

Platelet factor 4

Platelet factor 4 decreased

Platelet factor 4 increased

Platelet function test

Platelet function test abnormal

Platelet function test normal

Platelet glycoprotein gene mutation


Platelet maturation arrest

Platelet morphology

Platelet morphology abnormal

Platelet morphology normal

Platelet production decreased

Platelet storage pool deficiency

Platelet toxicity

Platelet-large cell ratio

Platelet-large cell ratio decreased

Platelet-large cell ratio increased

Plateletcrit

Plateletcrit abnormal

Plateletcrit decreased

Plateletcrit increased

Plateletcrit normal

Poikilocytosis

Polychromasia

Polychromic red blood cells present

Polyclonal B-cell lymphocytosis

Polycythaemia

Polycythaemia neonatorum

Polycythaemia vera

Polymorphonuclear chromatin clumping

Post transfusion purpura

Post transplant distal limb syndrome

Post transplant lymphoproliferative disorder

Post-anaphylaxis mast cell anergy

Post-depletion B-cell recovery

Postmastectomy lymphoedema syndrome

Postoperative lymphocele

Postsplenectomy syndrome

Precursor B-lymphoblastic lymphoma

Precursor B-lymphoblastic lymphoma recurrent

Precursor B-lymphoblastic lymphoma refractory

Precursor B-lymphoblastic lymphoma stage I

Precursor B-lymphoblastic lymphoma stage II

Precursor B-lymphoblastic lymphoma stage III

Precursor B-lymphoblastic lymphoma stage IV

Precursor T-lymphoblastic leukaemia acute

Precursor T-lymphoblastic lymphoma/leukaemia

Precursor T-lymphoblastic lymphoma/leukaemia recurrent

Precursor T-lymphoblastic lymphoma/leukaemia refractory

Precursor T-lymphoblastic lymphoma/leukaemia stage I

Precursor T-lymphoblastic lymphoma/leukaemia stage II

Precursor T-lymphoblastic lymphoma/leukaemia stage III

Precursor T-lymphoblastic lymphoma/leukaemia stage IV

Prekallikrein decreased

Prekallikrein increased

Prekallikrein test

Prekallikrein test abnormal

Prekallikrein test normal

Primary breast lymphoma

Primary cardiac lymphoma

Primary effusion lymphoma

Primary gastrointestinal follicular lymphoma

Primary mediastinal large B-cell lymphoma

Primary mediastinal large B-cell lymphoma recurrent

Primary mediastinal large B-cell lymphoma refractory

Primary mediastinal large B-cell lymphoma stage I

Primary mediastinal large B-cell lymphoma stage II

Primary mediastinal large B-cell lymphoma stage III

Primary mediastinal large B-cell lymphoma stage IV

Primary myelofibrosis

Proerythroblast count

Proerythroblast count abnormal

Proerythroblast count decreased

Proerythroblast count increased

Proerythroblast count normal

Prolymphocytic leukaemia

Promyelocyte count

Promyelocyte count decreased

Promyelocyte count increased

Protein C

Protein C decreased

Protein C deficiency

Protein C increased

Protein S

Protein S abnormal

Protein S decreased

Protein S deficiency

Protein S increased

Protein S normal

Protein deficiency anaemia

Prothrombin consumption time prolonged

Prothrombin consumption time shortened

Prothrombin fragment 1.2

Prothrombin fragment 1.2 increased

Prothrombin index

Prothrombin level

Prothrombin level abnormal

Prothrombin level decreased

Prothrombin level increased Prothrombin level normal

Prothrombin time

Prothrombin time abnormal

Prothrombin time normal

Prothrombin time prolonged

Prothrombin time ratio

Prothrombin time ratio abnormal

Prothrombin time ratio decreased

Prothrombin time ratio increased

Prothrombin time shortened

Pseudolymphoma

Pseudomononucleosis

Pulmonary eosinophilia

Pulmonary lymphangiectasia

Pulmonary nodular lymphoid hyperplasia


Punctate basophilia

Pure white cell aplasia
Purpura

Purpura fulminans

Purpura neonatal

Purpura non-thrombocytopenic

Purpura senile

Pyruvate kinase deficiency anaemia

Radiation leukopenia

Radiation-induced lymphocyte apoptosis

Red blood cell Heinz bodies present

Red blood cell abnormality

Red blood cell acanthocytes present

Red blood cell agglutination

Red blood cell agglutination present

Red blood cell analysis

Red blood cell analysis abnormal

Red blood cell analysis normal

Red blood cell anisocytes

Red blood cell anisocytes present

Red blood cell burr cells present

Red blood cell count

Red blood cell count abnormal

Red blood cell count decreased

Red blood cell count increased

Red blood cell count normal

Red blood cell elliptocytes present

Red blood cell enzymes abnormal

Red blood cell hyperchromic morphology

Red blood cell hyperchromic morphology present

Red blood cell hypochromic morphology present

Red blood cell macrocytes present

Red blood cell microcytes

Red blood cell microcytes absent

Red blood cell microcytes present

Red blood cell morphology

Red blood cell morphology abnormal

Red blood cell morphology normal

Red blood cell nucleated morphology

Red blood cell nucleated morphology present

Red blood cell poikilocytes

Red blood cell poikilocytes present

Red blood cell punctate basophilia present

Red blood cell rouleaux formation present

Red blood cell schistocytes

Red blood cell schistocytes present

Red blood cell sedimentation rate

Red blood cell sedimentation rate abnormal

Red blood cell sedimentation rate decreased

Red blood cell sedimentation rate increased Red blood cell sedimentation rate normal


Red blood cell sickled cells present

Red blood cell siderocytes present

Red blood cell spherocytes

Red blood cell spherocytes present

Red blood cell target cells present

Red blood cell vacuolisation

Red cell distribution width

Red cell distribution width abnormal

Red cell distribution width decreased

Red cell distribution width increased

Red cell distribution width normal

Red cell fragmentation syndrome

Refractory anaemia with an excess of blasts

Refractory anaemia with ringed sideroblasts

Refractory cytopenia with multilineage dysplasia

Refractory cytopenia with unilineage dysplasia

Renal lymphocele

Renal-limited thrombotic microangiopathy

Reticular cell count

Reticulocyte count

Reticulocyte count abnormal

Reticulocyte count decreased

Reticulocyte count increased

Reticulocyte count normal

Reticulocyte haemoglobin equivalent

Reticulocyte percentage

Reticulocyte percentage abnormal

Reticulocyte percentage decreased

Reticulocyte percentage increased

Reticulocyte percentage normal

Reticulocytopenia

Reticulocytosis

Reticuloendothelial dysfunction

Reticuloendothelial system stimulated

Retinopathy sickle cell

Retroperitoneal lymphadenopathy

Rhesus antibodies

Rhesus antibodies negative

Rhesus antibodies positive

Rhesus antigen

Rhesus antigen negative

Rhesus antigen positive

Rhesus haemolytic disease of newborn

Rhesus incompatibility

Richter's syndrome

Rosai-Dorfman syndrome

Rouleaux formation

Russell's viper venom time

Russell's viper venom time abnormal


Russell's viper venom time normal

Scan bone marrow

Scan bone marrow abnormal

Scan bone marrow normal

Scan lymph nodes

Scan spleen

Schistocytosis

Schumm's test

Schumm's test negative

Schumm's test positive

Secondary thrombocytosis

Septic coagulopathy

Serum colour abnormal

Severe fever with thrombocytopenia syndrome

Sezary cell count

Sezary cells increased

Shift to the left

Shift to the right

Shwachman-Diamond syndrome

Sickle cell anaemia

Sickle cell anaemia with crisis

Sickle cell disease

Sickle cell nephropathy

Sickle cell trait

Sideroblastic anaemia

Solitary epithelioid histiocytoma

Soluble fibrin monomer complex

Soluble fibrin monomer complex increased

Spherocytic anaemia

Spleen atrophy

Spleen congestion

Spleen contusion

Spleen disorder

Spleen follicular hyperplasia

Spleen ischaemia

Spleen malformation

Spleen procedural complication

Spleen scan abnormal

Spleen scan normal

Spleen tuberculosis

Splenic abscess

Splenic artery perforation

Splenic artery stenosis

Splenic artery thrombosis

Splenic calcification

Splenic candidiasis

Splenic cyst

Splenic embolism

Splenic fibrosis

Splenic granuloma

Splenic haematoma

Splenic haemorrhage

Splenic hamartoma

Splenic induration

Splenic infarction

Splenic infection

Splenic infection bacterial

Splenic infection fungal

Splenic infection helminthic


Splenic infection viral

Splenic injury

Splenic lesion

Splenic marginal zone lymphoma

Splenic marginal zone lymphoma recurrent

Splenic marginal zone lymphoma refractory

Splenic marginal zone lymphoma stage I

Splenic marginal zone lymphoma stage II

Splenic marginal zone lymphoma stage III

Splenic marginal zone lymphoma stage IV

Splenic necrosis

Splenic neoplasm malignancy unspecified

Splenic peliosis

Splenic rupture

Splenic thrombosis

Splenic varices

Splenic varices haemorrhage

Splenic vein occlusion

Splenic vein thrombosis

Splenitis

Splenomegaly

Splenorenal shunt

Splenosis

Spontaneous haematoma

Spontaneous haemorrhage

Spontaneous heparin-induced thrombocytopenia syndrome

Spur cell anaemia

Sticky platelet syndrome

Stomatocytes present

Stress polycythaemia

Subacute combined cord degeneration

Subcapsular splenic haematoma

Sulphaemoglobinaemia

Systemic mastocytosis

T-cell chronic lymphocytic leukaemia

T-cell lymphoma

T-cell lymphoma recurrent

T-cell lymphoma refractory

T-cell lymphoma stage I

T-cell lymphoma stage II

T-cell lymphoma stage III

T-cell lymphoma stage IV

T-cell prolymphocytic leukaemia

T-cell type acute leukaemia

T-cell unclassifiable lymphoma high grade

T-cell unclassifiable lymphoma low grade


T-lymphocyte count

T-lymphocyte count abnormal

T-lymphocyte count decreased

T-lymphocyte count increased

T-lymphocyte count normal

TEMPI syndrome

Thalassaemia

Thalassaemia alpha

Thalassaemia beta

Thalassaemia minor

Thalassaemia sickle cell

Thrombasthenia

Thrombin time

Thrombin time abnormal

Thrombin time normal

Thrombin time prolonged

Thrombin time shortened

Thrombin-antithrombin III complex

Thrombin-antithrombin III complex abnormal

Thrombin-antithrombin III complex decreased

Thrombin-antithrombin III complex increased

Thrombin-antithrombin III complex normal

Thrombocytopenia

Thrombocytopenia neonatal

Thrombocytopenia-absent radius syndrome

Thrombocytopenic purpura

Thrombocytosis

Thromboelastogram

Thrombopoietin level abnormal

Thrombotic microangiopathy

Thrombotic thrombocytopenic purpura

Thromboxane decreased

Thromboxane increased

Thymic cancer metastatic

Thymic cyst

Thymoma

Thymoma benign

Thymoma malignant

Thymoma malignant recurrent

Thymus abscess

Thymus disorder

Thymus enlargement

Thymus hypoplasia

Thyroid B-cell lymphoma

Transcobalamin deficiency

Transformation to acute myeloid leukaemia

Transfusion reaction

Transfusion-related alloimmune neutropenia

Traumatic ulcerative granuloma with stromal eosinophilia

Triple hit lymphoma

Trisomy 12

Tropical eosinophilia

Tropical sprue

Tuberculosis of intrathoracic lymph nodes

Tuberculosis of peripheral lymph nodes

Ultrasound spleen

Vaccination site lymphadenopathy

Vascular purpura

Venolymphatic malformation

Vitamin C deficiency

Von Willebrand's disease

Von Willebrand's factor activity abnormal

Von Willebrand's factor activity decreased

Von Willebrand's factor activity increased

Von Willebrand's factor activity normal

Von Willebrand's factor activity test

Von Willebrand's factor antibody

Von Willebrand's factor antibody positive

Von Willebrand's factor antigen abnormal

Von Willebrand's factor antigen decreased

Von Willebrand's factor antigen increased

Von Willebrand's factor antigen normal

Von Willebrand's factor antigen test

Von Willebrand's factor inhibition

Von Willebrand's factor multimers abnormal

Von Willebrand's factor multimers normal

Von Willebrand's factor multimers test

Waldenstrom's macroglobulinaemia

Waldenstrom's macroglobulinaemia recurrent

Waldenstrom's macroglobulinaemia refractory

Waldenstrom's macroglobulinaemia stage I

Waldenstrom's macroglobulinaemia stage II

Waldenstrom's macroglobulinaemia stage III

Waldenstrom's macroglobulinaemia stage IV

Warm type haemolytic anaemia

White blood cell agglutination present

White blood cell analysis

White blood cell analysis abnormal

White blood cell analysis normal

White blood cell count

White blood cell count abnormal

White blood cell count decreased

White blood cell count increased

White blood cell count normal

White blood cell disorder

White blood cell morphology

White blood cell morphology abnormal

White blood cell morphology normal

White clot in blood present

Wiskott-Aldrich syndrome

X-linked lymphoproliferative syndrome

Acquired C1 inhibitor deficiency

Acute generalised exanthematous pustulosis

Acute respiratory failure

Administration related reaction

Administration site dermatitis

Administration site eczema

Administration site hypersensitivity

Administration site photosensitivity reaction


Administration site rash

Administration site recall reaction

Administration site urticaria

Administration site vasculitis

Airway remodelling

Allergic bronchitis

HYPERSENSITIVITY

Allergic colitis

Allergic cough

Allergic cystitis

Allergic eosinophilia

Allergic gastroenteritis

Allergic hepatitis

Allergic keratitis

Allergic oedema

Allergic otitis externa

Allergic otitis media

Allergic pharyngitis

Allergic reaction to excipient

Allergic respiratory disease

Allergic respiratory symptom

Allergic sinusitis

Allergic stomatitis

Allergic transfusion reaction

Allergy alert test positive

Allergy test positive

Allergy to chemicals

Allergy to fermented products

Allergy to immunoglobulin therapy

Allergy to surgical sutures

Allergy to vaccine

Alpha tumour necrosis factor increased

Alveolitis

Anal eczema

Anaphylactic reaction

Anaphylactic shock

Anaphylactic transfusion reaction

Anaphylactoid reaction

Anaphylactoid shock

Anaphylaxis treatment

Angioedema

Anti-insulin antibody increased

Anti-insulin antibody positive

Anti-insulin receptor antibody increased

Anti-insulin receptor antibody positive

Anti-neutrophil cytoplasmic antibody positive vasculitis

Antiallergic therapy

Antibody test abnormal

Antibody test positive

Antiendomysial antibody positive

Application site dermatitis

Application site eczema

Application site hypersensitivity

Application site photosensitivity reaction

Application site rash

Application site recall reaction

Application site urticaria

Application site vasculitis

Arthritis allergic

Aspirin-exacerbated respiratory disease

Asthma

Asthma late onset

Asthma-chronic obstructive pulmonary disease overlap syndrome

Asthmatic crisis

Atopic cough

Atopy

Auricular swelling

Blepharitis allergic

Blister

Blister rupture

Blood immunoglobulin A abnormal

Blood immunoglobulin A increased

Blood immunoglobulin D increased

Blood immunoglobulin E abnormal

Blood immunoglobulin E increased

Blood immunoglobulin G abnormal

Blood immunoglobulin G increased

Blood immunoglobulin M abnormal

Blood immunoglobulin M increased

Bromoderma

Bronchial hyperreactivity

Bronchial oedema

Bronchospasm

Bullous haemorrhagic dermatosis

Bullous impetigo

Caffeine allergy

Capillaritis

Catheter site dermatitis

Catheter site eczema

Catheter site hypersensitivity

Catheter site rash

Catheter site urticaria

Catheter site vasculitis

Charcot-Leyden crystals

Cheilitis

Childhood asthma

Choking

Choking sensation

Chronic eosinophilic rhinosinusitis

Chronic hyperplastic eosinophilic sinusitis

Circulatory collapse

Circumoral oedema

Circumoral swelling

Complement factor C1 decreased

Complement factor C2 decreased

Complement factor C3 decreased

Complement factor C4 decreased


Complement factor decreased

Conjunctival oedema

Conjunctivitis

Conjunctivitis allergic

Contact stomatitis

Contrast media allergy

Contrast media reaction

Corneal exfoliation

Corneal oedema

Cough variant asthma

Cross sensitivity reaction

Cutaneous vasculitis

Cytokine increased

Cytokine release syndrome

Cytokine storm

Dennie-Morgan fold

Dermatitis

Dermatitis acneiform

Dermatitis allergic

Dermatitis atopic

Dermatitis bullous

Dermatitis contact

Dermatitis exfoliative

Dermatitis exfoliative generalised

Dermatitis herpetiformis

Dermatitis infected

Dermatitis psoriasiform

Device allergy

Dialysis membrane reaction

Distributive shock

Documented hypersensitivity to administered product

Drug eruption

Drug hypersensitivity

Drug provocation test

Drug reaction with eosinophilia and systemic symptoms

Ear swelling

Eczema

Eczema infantile

Eczema nummular

Eczema vaccinatum

Eczema vesicular

Eczema weeping

Encephalitis allergic

Encephalopathy allergic

Eosinophil count abnormal

Eosinophil count increased

Eosinophil percentage abnormal

Eosinophil percentage increased

Eosinophilia

Eosinophilia myalgia syndrome

Eosinophilic bronchitis

Eosinophilic granulomatosis with polyangiitis


Eosinophilic oesophagitis

Eosinophilic pneumonia

Eosinophilic pneumonia acute

Eosinophilic pneumonia chronic

Epidermal necrosis

Epidermolysis

Epidermolysis bullosa

Epiglottic oedema

Erythema

Erythema multiforme

Erythema nodosum

Exfoliative rash

Eye allergy

Eye oedema

Eye swelling

Eyelid oedema

Face oedema

Fixed eruption

Flushing

Gastrointestinal oedema

Generalised bullous fixed drug eruption

Generalised oedema

Genital rash

Genital swelling

Giant papillary conjunctivitis

Gingival oedema

Gingival swelling

Gleich's syndrome

HLA marker study positive

Haemolytic transfusion reaction

Haemorrhagic urticaria

Hand dermatitis

Henoch-Schonlein purpura

Henoch-Schonlein purpura nephritis

Heparin-induced thrombocytopenia

Human anti-hamster antibody increased

Human anti-hamster antibody positive

Hypersensitivity

Hypersensitivity myocarditis

Hypersensitivity pneumonitis

Hypersensitivity vasculitis

Idiopathic urticaria

Immediate post-injection reaction

Immune complex level increased

Immune thrombocytopenia

Immune tolerance induction

Immunoglobulins abnormal

Immunoglobulins increased

Immunology test abnormal

Implant site dermatitis

Implant site hypersensitivity

Implant site photosensitivity

Implant site rash

Implant site urticaria

Incision site dermatitis

Incision site rash

Infusion related hypersensitivity reaction


Infusion related reaction

Infusion site dermatitis

Infusion site eczema

Infusion site hypersensitivity

Infusion site photosensitivity reaction

Infusion site rash

Infusion site recall reaction

Infusion site urticaria

Infusion site vasculitis

Injection related reaction

Injection site dermatitis

Injection site eczema

Injection site hypersensitivity

Injection site panniculitis

Injection site photosensitivity reaction

Injection site rash

Injection site recall reaction

Injection site urticaria

Injection site vasculitis

Instillation site hypersensitivity

Instillation site rash

Instillation site urticaria

Interstitial granulomatous dermatitis

Interstitial lung disease

Intestinal angioedema

Iodine allergy

Kounis syndrome

Laryngeal dyspnoea

Laryngeal obstruction

Laryngeal oedema

Laryngitis allergic

Laryngospasm

Laryngotracheal oedema

Leukotriene increased

Limbal swelling

Lip exfoliation

Lip oedema

Lip swelling

Localised oedema

Macrophage inflammatory protein-1 alpha increased

Mast cell activation syndrome

Mast cell degranulation present

Mechanical urticaria

Medical device site dermatitis

Medical device site eczema

Medical device site hypersensitivity

Medical device site photosensitivity reaction

Medical device site rash

Medical device site recall reaction

Medical device site urticaria

Mesenteric panniculitis

Monocyte chemotactic protein-2 increased


Mouth swelling

Mouth ulceration

Mucocutaneous rash

Mucocutaneous ulceration

Mucosa vesicle

Mucosal erosion

Mucosal exfoliation

Mucosal necrosis

Mucosal ulceration

Multiple allergies

Nasal crease

Necrotising panniculitis

Nephritis allergic

Neurodermatitis

Neutralising antibodies positive

Nikolsky's sign

Nodular rash

Non-neutralising antibodies positive

Noninfective conjunctivitis

Nutritional supplement allergy

Occupational asthma

Occupational dermatitis

Oculomucocutaneous syndrome

Oculorespiratory syndrome

Oedema mouth

Oedema mucosal

Oral allergy syndrome

Oral mucosal exfoliation

Orbital oedema

Oropharyngeal blistering

Oropharyngeal oedema

Oropharyngeal spasm

Oropharyngeal swelling

Palatal oedema

Palatal swelling

Palisaded neutrophilic granulomatous dermatitis

Palpable purpura

Panniculitis

Pathergy reaction

Penile exfoliation

Penile oedema

Penile rash

Penile swelling

Perineal rash

Perioral dermatitis

Periorbital oedema

Periorbital swelling

Perivascular dermatitis

Pharyngeal oedema

Pharyngeal swelling

Photosensitivity reaction

Pneumonitis

Procedural shock

Prurigo

Pruritus

Pruritus allergic

Pulmonary eosinophilia

Radioallergosorbent test positive

Rash

Rash erythematous

Rash follicular

Rash macular

Rash maculo-papular

Rash maculovesicular

Rash morbilliform

Rash neonatal

Rash papulosquamous

Rash pruritic

Rash pustular

Rash rubelliform

Rash scarlatiniform

Rash vesicular

Reaction to azo-dyes

Reaction to colouring

Reaction to excipient

Reaction to food additive

Reaction to preservatives

Reactive airways dysfunction syndrome

Red man syndrome

Respiratory arrest

Respiratory distress

Respiratory failure

- ·

Respiratory tract oedema

Reversible airways obstruction

Rhinitis allergic

Rhinitis perennial

SJS-TEN overlap

Scleral oedema

Scleritis allergic

Scrotal dermatitis

Scrotal exfoliation

Scrotal oedema

Scrotal swelling

Seasonal allergy

Septal panniculitis

Serum sickness

Serum sickness-like reaction

Shock

Shock symptom

Skin erosion

Skin exfoliation

Skin necrosis

Skin oedema

Skin reaction

Skin swelling

Skin test positive

Sneezing

Solar urticaria

Solvent sensitivity

Status asthmaticus

Stevens-Johnson syndrome

Stoma site hypersensitivity

Stoma site rash

Stomatitis

Streptokinase antibody increased

Stridor

Suffocation feeling

Sunscreen sensitivity

Swelling face

Swelling of eyelid

Swollen tongue

Symmetrical drug-related intertriginous and flexural exanthema

Throat tightness

Tongue exfoliation

Tongue oedema

Toxic epidermal necrolysis

Toxic skin eruption

Tracheal obstruction

Tracheal oedema

Tracheostomy

Transplantation associated food allergy

Type I hypersensitivity

Type II hypersensitivity

Type III immune complex mediated reaction

Type IV hypersensitivity reaction

Upper airway obstruction

Urticaria

Urticaria cholinergic

Urticaria chronic

Urticaria contact

Urticaria papular

Urticaria physical

Urticaria pigmentosa

Urticaria vesiculosa

Urticarial dermatitis

Urticarial vasculitis

Vaccination site dermatitis

Vaccination site eczema

Vaccination site exfoliation

Vaccination site hypersensitivity

Vaccination site photosensitivity reaction

Vaccination site rash

Vaccination site recall reaction

Vaccination site urticaria

Vaccination site vasculitis

Vaccination site vesicles

Vaccine associated enhanced disease

Vaccine associated enhanced respiratory disease


Vaginal oedema

Vaginal ulceration

Vasculitic rash

Vernal keratoconjunctivitis

Vessel puncture site rash

Vessel puncture site vesicles

Visceral oedema Vulval eczema Vulval oedema Vulval ulceration

Vulvovaginal exfoliation Vulvovaginal rash Vulvovaginal swelling Vulvovaginal ulceration Vulvovaginitis allergic

Wheezing

MANIC SWITCH Hypomania

Mania

Manic symptom

NEUROLEPTIC MALIGNANT SYNDROME

Altered state of consciousness

Autonomic nervous system imbalance Blood creatine phosphokinase MM increased Blood creatine phosphokinase abnormal Blood creatine phosphokinase increased

Blood pressure abnormal Blood pressure decreased Blood pressure fluctuation Blood pressure increased Body temperature increased Cardiovascular insufficiency

Catatonia Coma

Confusional state

Consciousness fluctuating

Delirium

Depressed level of consciousness

Disorientation
Dyskinesia
Dyslalia
Dysphagia
Dystonia
Dystonic tremor

Extrapyramidal disorder

Fatigue

Freezing phenomenon Heart rate abnormal Heart rate increased Hyperhidrosis Hyperkinesia Hyperpyrexia Hypertension

Hyperthermia malignant

Hypertonia

Hyporesponsive to stimuli


Hypotension

Labile blood pressure
Labile hypertension

Loss of consciousness Malignant catatonia

Muscle enzyme increased

Muscle necrosis Muscle rigidity Muscular weakness

Myalgia Myoclonus

Myoglobin blood increased Myoglobin blood present Myoglobin urine present Myoglobinaemia Myoglobinuria

Necrotising myositis

Neuroleptic malignant syndrome

Oculogyric crisis Opisthotonus Palpitations Parkinson's disease Parkinsonian crisis Parkinsonian rest tremor

Parkinsonism

Pyrexia

Respiratory failure Resting tremor Rhabdomyolysis Salivary hypersecretion Serotonin syndrome Slow response to stimuli

Stupor Tachycardia Tremor

Unresponsive to stimuli Urinary retention

White blood cell count abnormal White blood cell count increased

Withdrawal catatonia

ORTHOSTATIC HYPOTENSION, DIZZINESS, AND SYNCOPE

Dizziness

Dizziness postural Hypotension

Orthostatic hypotension

Presyncope Syncope Amenorrhoea

PROLACTIN Amenorrho

Amenorrhoea-galactorrhoea syndrome


Anorgasmia Blood prolactin

Blood prolactin abnormal Blood prolactin increased Breast discharge

Breast discharge Breast enlargement Breast swelling Ejaculation disorder Erectile dysfunction

Female orgasmic disorder

Female sexual dysfunction

Galactorrhoea

Gynaecomastia

Hirsutism

Hyperprolactinaemia

Hypomenorrhoea

Lactation disorder

Libido decreased

Loss of libido

Male sexual dysfunction

Menstrual disorder

Menstruation delayed

Menstruation irregular

Oligomenorrhoea

Orgasm abnormal

Orgasmic sensation decreased

Prolactin-producing pituitary tumour

Sexual dysfunction

Cardiac arrest

Cardiac death

Cardiac fibrillation

Cardio-respiratory arrest

Electrocardiogram QT interval abnormal

Electrocardiogram QT prolonged

Electrocardiogram U wave inversion

Electrocardiogram U wave present

Electrocardiogram U-wave abnormality

Electrocardiogram repolarisation abnormality

Long QT syndrome

Long QT syndrome congenital

Loss of consciousness

Sudden cardiac death

Sudden death

Syncope

Torsade de pointes

Ventricular arrhythmia

Ventricular fibrillation

Ventricular flutter

Ventricular tachyarrhythmia

Ventricular tachycardia

Acute kidney injury

Anuria

Biopsy muscle abnormal

Blood calcium decreased

Blood creatine phosphokinase MM increased


Blood creatine phosphokinase abnormal

Blood creatine phosphokinase increased

Blood creatinine abnormal

Blood creatinine increased

Chromaturia

Chronic kidney disease

QT PROLONGATION

RHABDOMYOLYSIS AND CPK ELEVATION

Compartment syndrome

Creatinine renal clearance abnormal

Creatinine renal clearance decreased

Diaphragm muscle weakness

Electromyogram abnormal

End stage renal disease

Glomerular filtration rate abnormal

Glomerular filtration rate decreased

Haematoma muscle

Hypercreatininaemia

Hypocalcaemia

Muscle discomfort

Muscle disorder

Muscle enzyme increased

Muscle fatigue

Muscle haemorrhage

Muscle necrosis

Muscle rupture

Muscle strength abnormal

Muscular weakness

Musculoskeletal discomfort

Musculoskeletal disorder

Musculoskeletal pain

Musculoskeletal toxicity

Myalgia

Myalgia intercostal

Myoglobin blood increased

Myoglobin blood present

Myoglobin urine present

Myoglobinaemia

Myoglobinuria

Myopathy

Myopathy toxic

Myositis

Necrotising myositis

Oliguria

Renal failure

Renal impairment

Renal tubular necrosis

Rhabdomyolysis

Subacute kidney injury

Tendon discomfort

Thyrotoxic myopathy

1p36 deletion syndrome

2-Hydroxyglutaric aciduria

Acquired epileptic aphasia

Acute encephalitis with refractory, repetitive partial seizures


Alcoholic seizure

Alpers disease

Amygdalohippocampectomy

Aspartate-glutamate-transporter deficiency

Atonic seizures

Atypical benign partial epilepsy

SEIZURES

Aura

Automatism epileptic

Autonomic seizure

Baltic myoclonic epilepsy

Benign familial neonatal convulsions

Benign rolandic epilepsy

Biotinidase deficiency

CDKL5 deficiency disorder

CEC syndrome

CSWS syndrome

Change in seizure presentation

Clonic convulsion

Congenital bilateral perisylvian syndrome

Convulsion in childhood

Convulsions local

Convulsive threshold lowered

Corpus callosotomy

Deja vu

Double cortex syndrome

Dreamy state

Drop attacks

Drug withdrawal convulsions

Early infantile epileptic encephalopathy with burst-suppression

Eclampsia

Epilepsy

Epilepsy surgery

Epilepsy with myoclonic-atonic seizures

Epileptic aura

Epileptic psychosis

Faciobrachial dystonic seizure

Febrile convulsion

Febrile infection-related epilepsy syndrome

Foaming at mouth

Focal cortical resection

Focal dyscognitive seizures

Frontal lobe epilepsy

GM2 gangliosidosis

Gelastic seizure

Generalised onset non-motor seizure

Generalised tonic-clonic seizure

Glucose transporter type 1 deficiency syndrome

Grey matter heterotopia

Hemiconvulsion-hemiplegia-epilepsy syndrome


Hemimegalencephaly

Hyperglycaemic seizure

Hypocalcaemic seizure

Hypoglycaemic seizure

Hyponatraemic seizure

Idiopathic generalised epilepsy

Infantile spasms

Jeavons syndrome

Juvenile absence epilepsy

Juvenile myoclonic epilepsy

Lafora's myoclonic epilepsy Lennox-Gastaut syndrome Migraine-triggered seizure Molybdenum cofactor deficiency Multiple subpial transection

Myoclonic epilepsy

Myoclonic epilepsy and ragged-red fibres

Narcolepsy

Neonatal epileptic seizure

Neonatal seizure
Parietal lobe epilepsy
Partial seizures

Partial seizures with secondary generalisation

Petit mal epilepsy
Polymicrogyria
Post stroke epilepsy
Post stroke seizure
Post-traumatic epilepsy
Postictal headache
Postictal paralysis
Postictal psychosis
Postictal state

Preictal state Schizencephaly

Seizure

Seizure anoxic Seizure cluster

Seizure like phenomena Seizure prophylaxis

Severe myoclonic epilepsy of infancy

Simple partial seizures Status epilepticus

Sudden unexplained death in epilepsy

Temporal lobe epilepsy

Tongue biting

Tonic clonic movements

Tonic convulsion Tonic posturing Topectomy

Transient epileptic amnesia Tuberous sclerosis complex

Uncinate fits

SOMNOLENCE Fatigue

Hypersomnia Malaise Sedation

Sedation complication

Somnolence

SUICIDALITY Assisted suicide

Columbia suicide severity rating scale abnormal


Completed suicide
Depression suicidal
Intentional overdose

Intentional self-injury Poisoning deliberate Self-injurious ideation Suicidal behaviour Suicidal ideation Suicide attempt Suicide threat Suspected suicide

VTE (THROMBOTIC AND EMBOLIC EVENTS)

Aseptic cavernous sinus thrombosis

Axillary vein thrombosis

Suspected suicide attempt

Brachiocephalic vein occlusion

Brachiocephalic vein thrombosis Budd-Chiari syndrome Catheter management

Catheterisation venous

Cavernous sinus thrombosis Central venous catheterisation Cerebral venous sinus thrombosis

Cerebral venous thrombosis

Compression garment application

Deep vein thrombosis

Deep vein thrombosis postoperative

Embolism venous Hepatic vein embolism Hepatic vein occlusion Hepatic vein thrombosis

Homans' sign positive Iliac vein occlusion

Inferior vena cava syndrome

Inferior vena caval occlusion

Jugular vein embolism

Jugular vein occlusion

Jugular vein thrombosis

Mahler sign

May-Thurner syndrome

Mesenteric vein thrombosis

Mesenteric venous occlusion

Obstetrical pulmonary embolism

Obstructive shock

Ophthalmic vein thrombosis

Ovarian vein thrombosis

Paget-Schroetter syndrome

Pelvic venous thrombosis

Penile vein thrombosis

Peripheral vein occlusion

Peripheral vein thrombus extension

Phlebectomy

Portal vein cavernous transformation

Portal vein embolism

Portal vein occlusion

Portal vein thrombosis

Portosplenomesenteric venous thrombosis

Post procedural pulmonary embolism

Post thrombotic syndrome

Postoperative thrombosis

Postpartum venous thrombosis

Pulmonary embolism

Pulmonary infarction

Pulmonary microemboli

Pulmonary oil microembolism

Pulmonary thrombosis

Pulmonary vein occlusion

Pulmonary veno-occlusive disease

Pulmonary venous thrombosis

Renal vein embolism

Renal vein occlusion

Renal vein thrombosis

Retinal vein occlusion

Retinal vein thrombosis

SI QIII TIII pattern

Septic pulmonary embolism

Splenic vein occlusion

Splenic vein thrombosis

Subclavian vein occlusion

Subclavian vein thrombosis

Superior sagittal sinus thrombosis

Superior vena cava occlusion

Superior vena cava syndrome

Thrombophlebitis

Thrombophlebitis migrans

Thrombophlebitis neonatal

Thrombophlebitis superficial

Thrombosed varicose vein

Thrombosis corpora cavernosa

Transverse sinus thrombosis

Vascular graft

Vena cava embolism

Vena cava filter insertion

Vena cava filter removal

Vena cava thrombosis

Venogram abnormal

Venoocclusive disease

Venoocclusive liver disease

Venous angioplasty

Venous occlusion

Venous operation

Venous recanalisation

Venous repair

Venous stent insertion

Venous thrombosis

Venous thrombosis in pregnancy


Venous thrombosis limb

Venous thrombosis neonatal

Visceral venous thrombosis

## Appendix 5 List of Summary Tables

| am 4.4 | |
|---|---|
| CT-1.1 | Subject Disposition During Phase B (Randomized Subjects) |
| CT-1.2 | Subject Disposition During Phase B by ADT (Randomized Subjects) |
| CT-1.3 | Subject Disposition During Phase A (Enrolled Subjects) |
| CT-1.4 | Subject Disposition During Phase A Plus (Phase A Plus Sample) |
| CT-2.1 | Reasons for Discontinuation During Phase B (Randomized Subjects) |
| CT-2.2 | Reasons for Discontinuation During Phase B by ADT (Randomized Subjects) |
| CT-2.3 | Reasons for Discontinuation During Phase A (Enrolled Subjects) |
| CT-2.4 | Reasons for Discontinuation During Phase A Plus (Phase A Plus Sample) |
| CT-2.5 | Subject Completion Rates by Time During Phase B (Randomized Subjects) |
| CT-3.1.1.1 | Demographic Characteristics (Full Analysis Set) |
| CT-3.1.1.2 | Demographic Characteristics by ADT: Duloxetine (Full Analysis Set) |
| CT-3.1.1.3 | Demographic Characteristics by ADT: Escitalopram (Full Analysis Set) |
| CT-3.1.1.4 | Demographic Characteristics by ADT: Fluvoxamine (Full Analysis Set) |
| CT-3.1.1.5 | Demographic Characteristics by ADT: Milnacipran (Full Analysis Set) |
| CT-3.1.1.6 | Demographic Characteristics by ADT: Paroxetine (Full Analysis Set) |
| CT-3.1.1.7 | Demographic Characteristics by ADT: Sertraline (Full Analysis Set) |
| CT-3.1.1.8 | Demographic Characteristics by ADT: Venlafaxine (Full Analysis Set) |
| CT-3.1.2.1 | Demographic Characteristics (Safety Analysis Set) |
| CT-3.1.2.2 | Demographic Characteristics by ADT: Duloxetine (Safety Analysis Set) |
| CT-3.1.2.3 | Demographic Characteristics by ADT: Escitalopram (Safety Analysis Set) |
| CT-3.1.2.4 | Demographic Characteristics by ADT: Fluvoxamine (Safety Analysis Set) |
| CT-3.1.2.5 | Demographic Characteristics by ADT: Milnacipran (Safety Analysis Set) |
| CT-3.1.2.6 | Demographic Characteristics by ADT: Paroxetine (Safety Analysis Set) |
| CT-3.1.2.7 | Demographic Characteristics by ADT: Sertraline (Safety Analysis Set) |
| CT-3.1.2.8 | Demographic Characteristics by ADT: Venlafaxine (Safety Analysis Set) |
| CT-3.1.3 | Demographic Characteristics (Pharmacokinetic Analysis Set) |
| CT-3.1.4 | Demographic Characteristics (ADT Sample) |
| CT-3.1.5 | Demographic Characteristics (Phase A Plus Sample) |
| CT-3.2.1.1 | Baseline Disease Characteristics (Full Analysis Set) |
| CT-3.2.1.2 | Baseline Disease Characteristics by ADT: Duloxetine (Full Analysis Set) |
| CT-3.2.1.3 | Baseline Disease Characteristics by ADT: Escitalopram (Full Analysis Set) |
| CT-3.2.1.4 | Baseline Disease Characteristics by ADT: Fluvoxamine (Full Analysis Set) |
| CT-3.2.1.5 | Baseline Disease Characteristics by ADT: Milnacipran (Full Analysis Set) |
| CT-3.2.1.6 | Baseline Disease Characteristics by ADT: Paroxetine (Full Analysis Set) |
| CT-3.2.1.7 | Baseline Disease Characteristics by ADT: Sertraline (Full Analysis Set) |
| CT-3.2.1.8 | Baseline Disease Characteristics by ADT: Venlafaxine (Full Analysis Set) |
| CT-3.2.2.1 | Baseline Disease Characteristics (Safety Analysis Set) |
| CT-3.2.2.2 | Baseline Disease Characteristics by ADT: Duloxetine (Safety Analysis Set) |
| CT-3.2.2.3 | Baseline Disease Characteristics by ADT: Escitalopram (Safety Analysis Set) |
| CT-3.2.2.4 | Baseline Disease Characteristics by ADT: Fluvoxamine (Safety Analysis Set) |
| CT-3.2.2.5 | Baseline Disease Characteristics by ADT: Milnacipran (Safety Analysis Set) |
| CT-3.2.2.6 | Baseline Disease Characteristics by ADT: Paroxetine (Safety Analysis Set) |
| CT-3.2.2.7 | Baseline Disease Characteristics by ADT: Sertraline (Safety Analysis Set) |
| CT-3.2.2.8 | Baseline Disease Characteristics by ADT: Venlafaxine (Safety Analysis Set) |
| CT-3.2.4 | Baseline Disease Characteristics (ADT Sample) |

| CT-3.2.5 | Baseline Disease Characteristics (Phase A Plus Sample) |
|---|---|
| CT-4.1.1 | Concomitant Medications: Medications Taken Prior to Start of Study Therapy (Safety Analysis Set) |
| CT-4.1.2 | Concomitant Medications: Medications Taken During Phase A (Safety Analysis Set) |
| CT-4.1.3 | Concomitant Medications: Medications Taken During Phase B (Safety Analysis Set) |
| CT-4.1.4 | Concomitant Medications: Medications Taken Post Study Period (Safety Analysis Set) |
| CT-4.1.5 | Psychiatric Concomitant Medications: Medications Taken Prior to Start of Study<br>Therapy (Safety Analysis Set) |
| CT-4.1.6 | Psychiatric Concomitant Medications: Medications Taken During Phase A (Safety Analysis Set) |
| CT-4.1.7 | Psychiatric Concomitant Medications: Medications Taken During Phase B (Safety Analysis Set) |
| CT-4.1.8 | Psychiatric Concomitant Medications: Medications Taken Post Study Period (Safety Analysis Set) |
| CT-4.2.1 | Concomitant Medications: Medications Taken During Phase A (ADT Sample) |
| CT-4.2.2 | Concomitant Medications: Medications Taken During Phase A Plus (Phase A Plus Sample) |
| CT-4.2.3 | Psychiatric Concomitant Medications: Medications Taken During Phase A (ADT Sample) |
| CT-4.2.4 | Psychiatric Concomitant Medications: Medications Taken During Phase A Plus (Phase A Plus Sample) |
| CT-4.4.1 | Summary of Major Protocol Deviations by Center and Type of Deviation (Randomized Subjects) |
| CT-4.4.2 | Summary of Major Protocol Deviations by Center and Type of Deviation (Non-randomized Subjects) |
| CT-5.1.1 | Summary of Efficacy Results at Week 6 of the Double-blind Period (Phase B) (Full Analysis Set) |
| CT-5.2.1 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score - MMRM (Full Analysis Set) |
| CT-5.2.2 | Summary of Mean Change From Baseline to Phase A by Study Week in MADRS Total Score (ADT Sample) |
| CT-5.2.3 | Summary of Mean Change From Baseline to Phase A and Phase A+ by Study Week in MADRS Total Score (Phase A Plus Sample) |
| CT-5.3.1 | Summary of Proportion of Subjects With a MADRS Response During Phase B Relative to the Baseline (End of Phase A) - LOCF (Full Analysis Set) |
| CT-5.3.2 | Summary of Proportion of Subjects With a MADRS Response During Phase B Relative to the Baseline (End of Phase A) - OC (Full Analysis Set) |
| CT-5.4.1 | Summary of Proportion of Subjects With a MADRS Remission During Phase B Relative to the Baseline (End of Phase A) - LOCF (Full Analysis Set) |
| CT-5.4.2 | Summary of Proportion of Subjects With a MADRS Remission During Phase B Relative to the Baseline (End of Phase A) - OC (Full Analysis Set) |
| CT-5.5.1 | Summary of Proportion of Subjects With a CGI-I Improvement During Phase B Relative to the Baseline (End of Phase A) - LOCF (Full Analysis Set) |
| CT-5.5.2 | Summary of Proportion of Subjects With a CGI-I Improvement During Phase B Relative to the Baseline (End of Phase A) - OC (Full Analysis Set) |
| CT-5.6.1 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in CGI-S - MMRM (Full Analysis Set) |
| CT-5.6.2 | Summary of Mean Change From Baseline to Phase A by Study Week in CGI-S (ADT Sample) |
| CT-5.6.3 | Summary of Mean Change From Baseline to Phase A and Phase A+ by Study Week in CGI-S (Phase A Plus Sample) |
| CT-5.7.1 | Summary of Mean Change From Baseline (End of Phase A) to Phase B in HAM-D 17<br>Total Score - LOCF (Full Analysis Set) |
| CT-5.7.2 | Summary of Mean Change From Baseline (End of Phase A) to Phase B in HAM-D 17<br>Total Score - OC (Full Analysis Set) |

| CT-5.7.3 | Summary of Mean Change From Baseline to Phase A in HAM-D 17 Total Score (ADT Sample) |
|---|---|
| CT-5.7.4 | Summary of Mean Change From Baseline to Phase A and Phase A+ in HAM-D 17 Total Score (Phase A Plus Sample) |
| CT-5.8.1 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in SDS Scores - MMRM (Full Analysis Set) |
| CT-5.8.2 | Summary of Mean Change From Baseline to Phase A by Study Week in SDS Scores (ADT Sample) |
| CT-5.8.3 | Summary of Mean Change From Baseline to Phase A and Phase A+ by Study Week in SDS Scores (Phase A Plus Sample) |
| CT-5.9.1 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS-S Total Score - MMRM (Full Analysis Set) |
| CT-5.9.2 | Summary of Mean Change From Baseline to Phase A by Study Week in MADRS-S Total Score (ADT Sample) |
| CT-5.9.3 | Summary of Mean Change From Baseline to Phase A and Phase A+ by Study Week in MADRS-S Total Score (Phase A Plus Sample) |
| CT-5.10.1 | Summary of Mean CGI-I Score by Study Week in Phase B Relative to Baseline (End of Phase A) - LOCF (Full Analysis Set) |
| CT-5.10.2 | Summary of Mean CGI-I Score by Study Week in Phase B Relative to Baseline (End of Phase A) - OC (Full Analysis Set) |
| CT-5.11.1 | Sensitivity Analysis of MNAR Using Tipping Point Analysis in MADRS Total Score<br>Assume All Dropouts as MNAR (Full Analysis Set) |
| CT-5.11.2 | Sensitivity Analysis of MNAR Using Tipping Point Analysis in MADRS Total Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Full Analysis Set) |
| CT-5.11.3 | Sensitivity Analysis of MNAR Using Tipping Point Analysis in MADRS Total Score Dropout due to AE or LOE as MNAR (Full Analysis Set) |
| CT-5.11.4 | Sensitivity Analysis of MNAR Using Placebo Based Imputation in MADRS Total Score (Full Analysis Set) |
| CT-5.11.5 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score - MI Wilcoxon Rank Sum Test, MI Robust Regression (Full Analysis Set) |
| CT-5.11.6 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score - OC Wilcoxon Rank Sum Test, OC Robust Regression (Full Analysis Set) |
| CT-6.1.1 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by ADT: Duloxetine - MMRM (Full Analysis Set) |
| CT-6.1.2 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by ADT: Escitalopram - MMRM (Full Analysis Set) |
| CT-6.1.3 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by ADT: Fluvoxamine - MMRM (Full Analysis Set) |
| CT-6.1.4 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by ADT: Milnacipran - MMRM (Full Analysis Set) |
| CT-6.1.5 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by ADT: Paroxetine - MMRM (Full Analysis Set) |
| CT-6.1.6 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by ADT: Sertraline - MMRM (Full Analysis Set) |
| CT-6.1.7 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by ADT: Venlafaxine - MMRM (Full Analysis Set) |
| CT-6.2.1 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Gender: Male - MMRM (Full Analysis Set) |
| CT-6.2.2 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Gender: Female - MMRM (Full Analysis Set) |
| CT-6.3.1 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Age: <55 Years - MMRM (Full Analysis Set) |

CT-6.3.2 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Age: >=55 Years - MMRM (Full Analysis Set) CT-6.4.1 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Number of Previous Adequate Antidepressant Treatments: 1 Treatment - MMRM (Full Analysis Set) Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week CT-6.4.2 in MADRS Total Score by Number of Previous Adequate Antidepressant Treatments: 2 Treatments - MMRM (Full Analysis Set) CT-6.4.3 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Number of Previous Adequate Antidepressant Treatments: 3 Treatments - MMRM (Full Analysis Set) CT-6.5.1 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by DSM-5 Diagnosis: Single Episode - MMRM (Full Analysis CT-6.5.2 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by DSM-5 Diagnosis: Recurrent Episode - MMRM (Full CT-6.6.1 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Number of Previous Depressive Episodes: 1 Episode -MMRM (Full Analysis Set) CT-6.6.2 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Number of Previous Depressive Episodes: 2 Episodes -MMRM (Full Analysis Set) Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week CT-6.6.3 in MADRS Total Score by Number of Previous Depressive Episodes: 3 or more Episodes- MMRM (Full Analysis Set) CT-6.7.1 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Duration of Current Episode: <=Median - MMRM (Full Analysis Set) CT-6.7.2 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Duration of Current Episode: >Median - MMRM (Full Analysis Set) Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week CT-6.8.1 in MADRS Total Score by Baseline MADRS Total Score: <= Median - MMRM (Full Analysis Set) Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week CT-6.8.2 in MADRS Total Score by Baseline MADRS Total Score: >Median - MMRM (Full Analysis Set) CT-6.9.1 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Ultrashort-acting Sedative-hypnotic Drugs: Present - MMRM (Full Analysis Set) CT-6.9.2 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Ultrashort-acting Sedative-hypnotic Drugs: Absent - MMRM (Full Analysis Set) CT-6.10.1 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Baseline Weight: <= Median - MMRM (Full Analysis Set) CT-6.10.2 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Baseline Weight: >Median - MMRM (Full Analysis Set) Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week CT-6.11.1 in MADRS Total Score by Baseline BMI: <=Median - MMRM (Full Analysis Set) CT-6.11.2 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Baseline BMI: >Median - MMRM (Full Analysis Set) CT-6.12.1 Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by CYP2D6 Metabolism Status: IM - MMRM (Full Analysis Set)

| CT-6.12.2 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by CYP2D6 Metabolism Status: EM - MMRM (Full Analysis Set) |
|---|---|
| CT-6.13.1 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Impact of COVID-19 Pandemic: Subjects |
| CT-6.13.2 | Completed/Discontinued before 07APR2020 - MMRM (Full Analysis Set) Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score by Impact of COVID-19 Pandemic: Subjects Completed/Discontinued on or after 07APR2020 - MMRM (Full Analysis Set) |
| CF-1 | Mean Change From Baseline (End of Phase A) to Phase B by Study Week in MADRS Total Score - MMRM (Full Analysis Set) |
| CT-7.1.1 | Extent of Exposure to Study Medication During Phase B (Safety Analysis Set) |
| CT-7.1.2 | Extent of Exposure to ADT During Phase B (Safety Analysis Set) |
| CT-7.1.3 | Extent of Exposure to ADT During Phase A (ADT Sample) |
| CT-7.1.4 | Extent of Exposure to ADT During Phase A Plus (Phase A Plus Sample) |
| CT-7.1.5 | Average Daily Dose ADT During Phase B (Safety Analysis Set) |
| CT-7.2 | Summary of Treatment Compliance (Full Analysis Set) |
| CT-8.1 | Adverse Events During Phase B (All Causalities) (Safety Analysis Set) |
| CT-8.2.1 | Incidence of TEAEs During Phase B by MedDRA System Organ Class and Preferred Term (Safety Analysis Set) |
| CT-8.2.2 | Incidence of Drug-related TEAEs During Phase B by MedDRA System Organ Class and Preferred Term (Safety Analysis Set) |
| CT-8.3.1 | Incidence of TEAEs During Phase B by MedDRA System Organ Class, Preferred Term and Severity (Safety Analysis Set) |
| CT-8.3.2 | Incidence of Drug-related TEAEs During Phase B by MedDRA System Organ Class, Preferred Term and Severity (Safety Analysis Set) |
| CT-8.4.1 | Incidence of Deaths due to TEAEs During Phase B by MedDRA System Organ Class and Preferred Term (Safety Analysis Set) |
| CT-8.4.2 | Incidence of Deaths due to Drug-related TEAEs During Phase B by MedDRA System Organ Class and Preferred Term (Safety Analysis Set) |
| CT-8.5.1 | Incidence of Serious TEAEs During Phase B by MedDRA System Organ Class and Preferred Term (Safety Analysis Set) |
| CT-8.5.2 | Incidence of Serious Drug-related TEAEs During Phase B by MedDRA System Organ Class and Preferred Term (Safety Analysis Set) |
| CT-8.6.1 | Incidence of TEAEs Resulting in Discontinuation of IMP During Phase B by MedDRA System Organ Class and Preferred Term (Safety Analysis Set) |
| CT-8.6.2 | Incidence of Drug-related TEAEs Resulting in Discontinuation of IMP During Phase B by MedDRA System Organ Class and Preferred Term (Safety Analysis Set) |
| CT-8.7.1 | Incidence of TEAEs During Phase B of at Least 2% in Any Brexpiprazole Group and Greater Than Placebo by MedDRA System Organ Class and Preferred Term (Safety Analysis Set) |
| CT-8.7.2 | Incidence of Drug-related TEAEs During Phase B of at Least 2% in Any Brexpiprazole Group and Greater Than Placebo by MedDRA System Organ Class and Preferred Term (Safety Analysis Set) |
| CT-8.8.1 | Incidence of TEAEs During Phase B by MedDRA System Organ Class, Preferred Term and Time to First Onset (Safety Analysis Set) |
| CT-8.8.2 | Incidence of Drug-related TEAEs During Phase B by MedDRA System Organ Class, Preferred Term and Time to First Onset (Safety Analysis Set) |
| CT-8.9.1 | Incidence of TEAEs for EPS (Safety Analysis Set) |
| CT-8.9.2 | Incidence of TEAEs During Phase B for Neuroleptic Malignant Syndrome (Safety Analysis Set) |
| CT-8.9.3 | Incidence of TEAEs During Phase B for Rhabdomyolysis and CPK Elevation (Safety Analysis Set) |
| CT-8.9.4 | Incidence of TEAEs During Phase B for Seizures (Safety Analysis Set) |

| CT-8.9.5 | Incidence of TEAEs During Phase B for Orthostatic Hypotension, Dizziness, and Syncope (Safety Analysis Set) |
|---|---|
| CT-8.9.6 | Incidence of TEAEs During Phase B for Suicidality (Safety Analysis Set) |
| CT-8.9.7 | Incidence of TEAEs During Phase B for Somnolence (Safety Analysis Set) |
| CT-8.9.8 | Incidence of TEAEs During Phase B for Hypersensitivity (Safety Analysis Set) |
| CT-8.9.9 | Incidence of TEAEs During Phase B for VTE (Thrombotic and Embolic Events) (Safety |
| | Analysis Set) |
| CT-8.9.10 | Incidence of TEAEs During Phase B for Haematopoietic/Leukopenia (Safety Analysis Set) |
| CT-8.9.11 | Incidence of TEAEs During Phase B for Effect on Glucose (Safety Analysis Set) |
| CT-8.9.12 | Incidence of TEAEs During Phase B for Effect on Lipids (Safety Analysis Set) |
| CT-8.9.13 | Incidence of TEAEs During Phase B for Effect on Weight (Safety Analysis Set) |
| CT-8.9.14 | Incidence of TEAEs During Phase B for QT Prolongation (Safety Analysis Set) |
| CT-8.9.15 | Incidence of TEAEs During Phase B for Manic Switch (Safety Analysis Set) |
| CT-8.9.16 | Incidence of TEAEs During Phase B for Effect on Prolactin (Safety Analysis Set) |
| CT-8.10.1 | Incidence of TEAEs During Phase B by MedDRA System Organ Class and Preferred |
| 0.10.1 | Term, by ADT (Safety Analysis Set) |
| CT-8.10.2 | Incidence of TEAEs During Phase B by MedDRA System Organ Class and Preferred Term, by Gender (Safety Analysis Set) |
| CT-8.10.3 | Incidence of TEAEs During Phase B by MedDRA System Organ Class and Preferred |
| | Term, by Age (Safety Analysis Set) |
| CT-8.10.4 | Incidence of TEAEs During Phase B by MedDRA System Organ Class and Preferred |
| | Term, by CYP2D6 Metabolism Status (Safety Analysis Set) |
| CT-8.10.5 | Incidence of TEAEs During Phase B by MedDRA System Organ Class and Preferred Term, by Impact of COVID-19 Pandemic (Safety Analysis Set) |
| CT-8.11.1 | Incidence of TEAEs During Phase A by MedDRA System Organ Class and Preferred |
| CT 0 11 2 | Term (ADT Sample) |
| CT-8.11.2 | Incidence of TEAEs During Phase A Plus by MedDRA System Organ Class and Preferred Term (Phase A Plus Sample) |
| CT-9.1.1 | Listing of Deaths During Phase B |
| CT-9.1.2 | Listing of Deaths During Phase A and Phase A Plus |
| CT-9.2.1 | Listing of Serious Adverse Events During Phase B |
| CT-9.2.2 | Listing of Serious Adverse Events During Phase A and Phase A Plus |
| CT-9.2.2<br>CT-9.3.1 | Listing of Discontinuation of IMP due to Adverse Events During Phase B |
| CT-9.3.1<br>CT-9.3.2 | Listing of Discontinuation of IMP due to Adverse Events During Phase A and Phase A Listing of Discontinuation of IMP due to Adverse Events During Phase A and Phase A |
| | Plus |
| CT-10.1.1 | Mean Change From Baseline (End of Phase A) in Clinical Laboratory Test Results -<br>Serum Chemistry (Safety Analysis Set) |
| CT-10.1.2 | Mean Change From Baseline (End of Phase A) in Clinical Laboratory Test Results -<br>Hematology (Safety Analysis Set) |
| CT-10.1.3 | Mean Change From Baseline (End of Phase A) in Clinical Laboratory Test Results - Urinalysis (Safety Analysis Set) |
| CT-10.1.4 | Mean Change From Baseline (End of Phase A) in Clinical Laboratory Test Results - |
| | Prolactin, by Gender (Safety Analysis Set) |
| CT-10.1.5 | Mean Change From Baseline (End of Phase A) in Clinical Laboratory Test Results - Other Tests (Safety Analysis Set) |
| CT-10.2.1 | Shift Tables of Clinical Laboratory Test Results - Serum Chemistry (Safety Analysis Set) |
| CT-10.2.2 | Shift Tables of Clinical Laboratory Test Results - Hematology (Safety Analysis Set) |
| CT-10.2.3 | Shift Tables of Clinical Laboratory Test Results - Urinalysis 1 (Safety Analysis Set) |
| CT-10.2.4 | Shift Tables of Clinical Laboratory Test Results - Urinalysis 2 (Safety Analysis Set) |
| C1 10.2.T | onite radies of Chinear Eadoratory Test results - Officiry 5152 (Safety Findiysis Set) |

| CT-10.2.5 | Shift Tables of Clinical Laboratory Test Results - Prolactin, by Gender (Safety Analysis Set) |
|---|---|
| CT-10.2.6 | Shift Tables of Clinical Laboratory Test Results - Other Tests (Safety Analysis Set) |
| CT-10.3.1 | Incidence of Laboratory Test Values With Potential Clinical Relevance During Phase B (Safety Analysis Set) |
| CT-10.3.2 | Listing of Laboratory Test Values With Potential Clinical Relevance During Phase B by Subject (Safety Analysis Set) |
| CT-10.4.1 | Incidence of Potential Hy's Law Cases During Phase B (Safety Analysis Set) |
| CT-10.4.2 | Listing of Potential Hy's Law Cases During Phase B (Safety Analysis Set) |
| CT-10.5.1 | Incidence of Laboratory Test Values With Potential Clinical Relevance During Phase B - Prolactin (Safety Analysis Set) |
| CT-10.5.2 | Listing of Laboratory Test Values With Potential Clinical Relevance During Phase B - Prolactin (Safety Analysis Set) |
| CT-10.6.1 | Incidence of Treatment-emergent Significant Change in Lipids During Phase B (Safety Analysis Set) |
| CT-10.6.2 | Listing of Treatment-emergent Significant Change in Lipids During Phase B (Safety Analysis Set) |
| CT-10.7.1 | Incidence of Treatment-emergent Significant Change in Glucose During Phase B (Safety Analysis Set) |
| CT-10.7.2 | Listing of Treatment-emergent Significant Change in Glucose During Phase B (Safety Analysis Set) |
| CT-10.8.1 | Incidence of Treatment-emergent Metabolic Syndrome During Phase B (Safety Analysis Set) |
| CT-10.8.2 | Listing of Treatment-emergent Metabolic Syndrome During Phase B (Safety Analysis Set) |
| CT-10.9.1 | Mean Change From Baseline in Clinical Laboratory Test Results During Phase A - Serum Chemistry (ADT Sample) |
| CT-10.9.2 | Mean Change From Baseline in Clinical Laboratory Test Results During Phase A - Hematology (ADT Sample) |
| CT-10.9.3 | Mean Change From Baseline in Clinical Laboratory Test Results During Phase A - Urinalysis (ADT Sample) |
| CT-10.9.4 | Mean Change From Baseline in Clinical Laboratory Test Results During Phase A - Prolactin, by Gender (ADT Sample) |
| CT-10.9.5 | Mean Change From Baseline in Clinical Laboratory Test Results During Phase A - Other Tests (ADT Sample) |
| CT-10.10.1 | Mean Change From Baseline in Clinical Laboratory Test Results During Phase A and Phase A+ - Serum Chemistry (Phase A Plus Sample) |
| CT-10.10.2 | Mean Change From Baseline in Clinical Laboratory Test Results During Phase A and Phase A+ - Hematology (Phase A Plus Sample) |
| CT-10.10.3 | Mean Change From Baseline in Clinical Laboratory Test Results During Phase A and Phase A+ - Urinalysis (Phase A Plus Sample) |
| CT-10.10.4 | Mean Change From Baseline in Clinical Laboratory Test Results During Phase A and Phase A+ - Prolactin, by Gender (Phase A Plus Sample) |
| CT-10.10.5 | Mean Change From Baseline in Clinical Laboratory Test Results During Phase A and Phase A+ - Other Tests (Phase A Plus Sample) |
| CT-10.11.1 | Listing of Laboratory Test Values With Potential Clinical Relevance During Phase A by Subject (ADT Sample) |
| CT-10.11.2 | Listing of Laboratory Test Values With Potential Clinical Relevance During Phase A and Phase A+ (Phase A Plus Sample) |
| CT-11.1 | Mean Change From Baseline (End of Phase A) in Vital Signs During Phase B (Safety Analysis Set) |
| CT-11.2 | Incidence of Potentially Clinically Relevant Abnormalities in Vital Signs During Phase B (Safety Analysis Set) |
| CT-11.3 | Listing of Potentially Clinically Relevant Abnormalities in Vital Signs During Phase B (Safety Analysis Set) |

| CT-11.4 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in Body Weight (kg) (Safety Analysis Set) |
|---|---|
| CT-11.5 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in Waist Circumference (cm) (Safety Analysis Set) |
| CT-11.6 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in BMI (kg/m^2) (Safety Analysis Set) |
| CT-11.7 | Incidence of Potentially Clinically Relevant Weight Gain or Loss by Baseline BMI (Safety Analysis Set) |
| CT-11.8 | Mean Change From Baseline in Vital Signs During Phase A (ADT Sample) |
| CT-11.9 | Mean Change From Baseline in Vital Signs During Phase A and Phase A+ (Phase A Plus Sample) |
| CT-11.10 | Listing of Potentially Clinically Relevant Abnormalities in Vital Signs During Phase A (ADT Sample) |
| CT-11.11 | Listing of Potentially Clinically Relevant Abnormalities in Vital Signs During Phase A and Phase A+ (Phase A Plus Sample) |
| CT-12.1 | Mean Change From Baseline (End of Phase A) in ECG Results During Phase B (Safety Analysis Set) |
| CT-12.2 | Shift Tables of ECG (Safety Analysis Set) |
| CT-12.3 | Incidence of Categorical Changes in QT/QTc During Phase B (Safety Analysis Set) |
| CT-12.4 | Incidence of Potentially Clinically Relevant Abnormalities in ECG Evaluations During Phase B (Safety Analysis Set) |
| CT-12.5 | Listing of Potentially Clinically Relevant Abnormalities in ECG Evaluations During Phase B (Safety Analysis Set) |
| CT-12.6 | Mean Change From Baseline in ECG Results During Phase A (ADT Sample) |
| CT-12.7 | Mean Change From Baseline in ECG Results During Phase A and Phase A+ (Phase A Plus Sample) |
| CT-12.8 | Listing of Potentially Clinically Relevant Abnormalities in ECG Evaluations During Phase A (ADT Sample) |
| CT-12.9 | Listing of Potentially Clinically Relevant Abnormalities in ECG Evaluations During Phase A and Phase A+ (Phase A Plus Sample) |
| CT-13.1 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in DIEPSS (Safety Analysis Set) |
| CT-13.2 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in AIMS Total Score and Item Scores 8, 9 and 10 (Safety Analysis Set) |
| CT-13.3 | Summary of Mean Change From Baseline (End of Phase A) to Phase B by Study Week in BARS, Global Clinical Assessment of Akathisia (Safety Analysis Set) |
| CT-13.4 | Summary of Mean Change From Baseline (End of Phase A) to Phase A+ by Study Week in DIEPSS (Phase A Plus Sample) |
| CT-13.5 | Summary of Mean Change From Baseline (End of Phase A) to Phase A+ by Study Week in AIMS Total Score and Item Scores 8, 9 and 10 (Phase A Plus Sample) |
| CT-13.6 | Summary of Mean Change From Baseline (End of Phase A) to Phase A+ by Study Week in BARS, Global Clinical Assessment of Akathisia (Phase A Plus Sample) |
| CT-14.1 | C-SSRS During Phase B, Suicidality (Safety Analysis Set) |
| CT-14.2 | C-SSRS During Phase B, Suicidal Behavior by Type (Safety Analysis Set) |
| CT-14.3 | C-SSRS During Phase B, Suicidal Ideation by Type (Safety Analysis Set) |
| CT-14.4 | C-SSRS During Phase B, Treatment Emergent Suicidal Behavior and Ideation (Safety Analysis Set) |
| CT-14.5 | C-SSRS - Listing of Treatment-emergent Suicidal Ideation During Phase B (Safety Analysis Set) |
| CT-14.6 | C-SSRS - Listing of Treatment-emergent Suicidal Behavior During Phase B (Safety Analysis Set) |
| CT-14.7 | C-SSRS - Listing of Treatment-emergent Serious Ideation During Phase B (Safety Analysis Set) |
| CT-14.8 | C-SSRS - Listing of Worsening Suicidal Ideation During Phase B (Safety Analysis Set) |

| CT 14.0 | C CCDC During Diago A Cuisidal Daharian by Tuna (ADT Canada) |
|---|---|
| CT-14.9 | C-SSRS During Phase A, Suicidal Behavior by Type (ADT Sample) |
| CT-14.10 | C-SSRS During Phase A, Suicidal Ideation by Type (ADT Sample) |
| CT-14.11 | C-SSRS During Phase A+, Suicidal Behavior by Type (Phase A Plus Sample) |
| CT-14.12 | C-SSRS During Phase A+, Suicidal Ideation by Type (Phase A Plus Sample) |
| PKT-1 | Individual Subject and Summary of Brexpiprazole Plasma Concentrations Following 1 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis |
| PKT-2 | Set) Individual Subject and Summary of Brexpiprazole Plasma Concentrations Following 2 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKT-3 | Summary of Brexpiprazole Plasma Concentrations for Each CYP2D6 Phenotype Following 1 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKT-4 | Summary of Brexpiprazole Plasma Concentrations for Each CYP2D6 Phenotype Following 2 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKT-5 | Summary of Brexpiprazole Plasma Concentrations for Each Requisite Concomitant Medication Following 1 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKT-6 | Summary of Brexpiprazole Plasma Concentrations for Each Requisite Concomitant Medication Following 2 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKF-1 | Mean (SD) and Scatter Plots of Brexpiprazole Plasma Concentrations Following 1 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis |
| PKF-2 | Set) Mean (SD) and Scatter Plots of Brexpiprazole Plasma Concentrations Following 2 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis |
| PKF-3 | Set) Mean (SD) and Scatter Plots of Brexpiprazole Plasma Concentrations for Each CYP2D6 Phenotype Following 1 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKF-4 | Mean (SD) and Scatter Plots of Brexpiprazole Plasma Concentrations for Each CYP2D6 Phenotype Following 2 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKF-5 | Mean (SD) and Scatter Plots of Brexpiprazole Plasma Concentrations for Each Requisite Concomitant Medication Following 1 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKF-6 | Mean (SD) and Scatter Plots of Brexpiprazole Plasma Concentrations for Each Requisite Concomitant Medication Following 2 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKF-7 | Scatter Plot of Brexpiprazole Plasma Concentrations Following 1 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKF-8 | Scatter Plot of Brexpiprazole Plasma Concentrations Following 2 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKF-9 | Scatter Plot of Brexpiprazole Plasma Concentrations for Each CYP2D6 Phenotype Following 1 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKF-10 | Scatter Plot of Brexpiprazole Plasma Concentrations for Each CYP2D6 Phenotype Following 2 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |
| PKF-11 | Scatter Plot of Brexpiprazole Plasma Concentrations for Each Requisite Concomitant Medication Following 1 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set) |

## Protocol 331-102-00058

PKF-12 Scatter Plot of Brexpiprazole Plasma Concentrations for Each Requisite Concomitant Medication Following 2 mg/day Doses of Brexpiprazole at Week 3 During Phase B (Pharmacokinetic Analysis Set)

## Appendix 6 List of Subject Data Listings

| A TO 1 1 | A.1. F. (P. 1. 10.11. () |
|---|---|
| AE-1.1 | Adverse Events (Randomized Subjects) |
| AE-1.2 | Adverse Events (Non-randomized Subjects) |
| DEMOG-1.1 | Demographic Characteristics (Randomized Subjects) |
| DEMOG-1.2 | Demographic Characteristics (Non-randomized Subjects) |
| DREAS-1.1 | Discontinued Subjects and Reason for Discontinuation (Randomized Subjects) |
| DREAS-1.2 | Discontinued Subjects and Reason for Discontinuation (Non-randomized Subjects) |
| LAB-1.1 | Laboratory Test Results: Serum Chemistry (Randomized Subjects) |
| LAB-1.2 | Laboratory Test Results: Serum Chemistry (Non-randomized Subjects) |
| LAB-2.1 | Laboratory Test Results: Hematology (Randomized Subjects) |
| LAB-2.2 | Laboratory Test Results: Hematology (Non-randomized Subjects) |
| LAB-3.1 | Laboratory Test Results: Urinalysis (Randomized Subjects) |
| LAB-3.2 | Laboratory Test Results: Urinalysis (Non-randomized Subjects) |
| LAB-4.1 | Laboratory Test Results: Other Laboratory Tests (Randomized Subjects) |
| LAB-4.2 | Laboratory Test Results: Other Laboratory Tests (Non-randomized Subjects) |
| LAB-5.1 | Pregnancy Test (Randomized Subjects) |
| LAB-5.2 | Pregnancy Test (Non-randomized Subjects) |
| EFF-1.1 | Montgomery Asberg Depression Rating Scale (MADRS) (Randomized Subjects) |
| EFF-1.2 | Montgomery Asberg Depression Rating Scale (MADRS) (Non-randomized Subjects) |
| EFF-2.1 | Clinical Global Impression - Severity of Illness (CGI-S) (Randomized Subjects) |
| EFF-2.2 | Clinical Global Impression - Severity of Illness (CGI-S) (Non-randomized Subjects) |
| EFF-3.1 | Clinical Global Impression - Improvement (CGI-I) (Randomized Subjects) |
| EFF-3.2 | Clinical Global Impression - Improvement (CGI-I) (Non-randomized Subjects) |
| EFF-4.1 | Hamilton Depression Rating Scale (HAM-D) (Randomized Subjects) |
| EFF-4.2 | Hamilton Depression Rating Scale (HAM-D) (Non-randomized Subjects) |
| EFF-5.1 | Montgomery Asberg Depression Rating Scale Self-assessment (MADRS-S) (Randomized Subjects) |
| EFF-5.2 | Montgomery Asberg Depression Rating Scale Self-assessment (MADRS-S) (Non-randomized Subjects) |
| EFF-6.1 | Sheehan Disability Scale (SDS) (Randomized Subjects) |
| EFF-6.2 | Sheehan Disability Scale (SDS) (Non-randomized Subjects) |
| PDATA-1.1 | Inclusion and Exclusion Criteria (Randomized Subjects) |
| PDATA-1.2 | Inclusion and Exclusion Criteria (Non-randomized Subjects) |
| PDATA-2 | Subject Randomization List (Randomized Subjects) |
| PDATA-3.1 | Study Completion Status and Reasons for Discontinuation (Randomized Subjects) |
| PDATA-3.2 | Study Completion Status and Reasons for Discontinuation (Non-randomized Subjects) |
| PDATA-4.1.1 | Prior and Concomitant Medications (Randomized Subjects) |
| PDATA-4.1.2 | Prior and Concomitant Medications (Non-randomized Subjects) |
| PDATA-4.2.1 | Prior Medication for Current Major Depressive Episode (Antidepressant) |
| <b>.</b> | (Randomized Subjects) |
| PDATA-4.2.2 | Prior Medication for Current Major Depressive Episode (Antidepressant) (Non- |
| | randomized Subjects) |
| PDATA-4.3.1 | Prior and Concomitant Therapy (Randomized Subjects) |
| PDATA-4.3.2 | Prior and Concomitant Therapy (Non-randomized Subjects) |
| PDATA-4.4.1 | Prior Therapy for Current Major Depressive Episode (Psychotherapy/Somatic Therapy) (Randomized Subjects) |

| PDATA-4.4.2 | Prior Therapy for Current Major Depressive Episode (Psychotherapy/Somatic Therapy) (Non-randomized Subjects) |
|---|---|
| PDATA-5.1 | Medical History (Randomized Subjects) |
| PDATA-5.2 | Medical History (Non-randomized Subjects) |
| PDATA-6.1 | Psychiatric Evaluation of Depression (Randomized Subjects) |
| PDATA-6.2 | Psychiatric Evaluation of Depression (Non-randomized Subjects) |
| PDATA-7.1 | Physical Examination (Randomized Subjects) |
| PDATA-7.2 | Physical Examination (Non-randomized Subjects) |
| PDATA-8.1 | Vital Signs (Randomized Subjects) |
| PDATA-8.2 | Vital Signs (Non-randomized Subjects) |
| PDATA-9.1 | Electrocardiogram Results (Randomized Subjects) |
| PDATA-9.2 | Electrocardiogram Results (Non-randomized Subjects) |
| PDATA-10.1.1 | Columbia-Suicide Severity Rating Scale (C-SSRS) - Suicidal Ideation and Intensity (Randomized Subjects) |
| PDATA-10.1.2 | Columbia-Suicide Severity Rating Scale (C-SSRS) - Suicidal Behavior (Randomized Subjects) |
| PDATA-10.1.3 | Columbia-Suicide Severity Rating Scale (C-SSRS) - Actual Attempts (Randomized Subjects) |
| PDATA-10.2.1 | Columbia-Suicide Severity Rating Scale (C-SSRS) - Suicidal Ideation and Intensity (Non-randomized Subjects) |
| PDATA-10.2.2 | Columbia-Suicide Severity Rating Scale (C-SSRS) - Suicidal Behavior (Non-randomized Subjects) |
| PDATA-10.2.3 | Columbia-Suicide Severity Rating Scale (C-SSRS) - Actual Attempts (Non-randomized Subjects) |
| PDATA-11.1 | Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) (Randomized Subjects) |
| PDATA-11.2 | Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) (Non-randomized Subjects) |
| PDATA-12.1 | Barnes Akathisia Rating Scale (BARS) (Randomized Subjects) |
| PDATA-12.2 | Barnes Akathisia Rating Scale (BARS) (Non-randomized Subjects) |
| PDATA-13.1 | Abnormal Involuntary Movement Scale (AIMS) (Randomized Subjects) |
| PDATA-13.2 | Abnormal Involuntary Movement Scale (AIMS) (Non-randomized Subjects) |
| PDATA-14 | Pharmacokinetic Blood Draw Time (Randomized Subjects) |
| PDATA-15.1 | CYP2D6 Genetic Test (Randomized Subjects) |
| PDATA-16.1 | Blood Draw Time for DNA Storage and Biomarker (Randomized Subjects) |
| PDATA-16.2 | Blood Draw Time for DNA Storage and Biomarker (Non-randomized Subjects) |
| PDATA-17.1 | Post-treatment Follow-up (Randomized Subjects) |
| PDATA-17.2 | Post-treatment Follow-up (Non-randomized Subjects) |
| PDATA-18 | Screening Failures |
| PDEV-1.1 | Major Protocol Deviations by Type of Deviation (Randomized Subjects) |
| PDEV-1.2 | Major Protocol Deviations by Type of Deviation (Non-randomized Subjects) |
| SMED-1.1 | Study Medication Administration (Randomized Subjects) |
| SMED-1.2 | Study Medication Administration - Antidepressant (Randomized Subjects) |
| SMED-2.1 | Study Medication Administration (Non-randomized Subjects) |
| SMED-2.2 | Study Medication Administration - Antidepressant (Non-randomized Subjects) |
| SMED-3.1 | Study Medication Compliance (Randomized Subjects) |
| SUBEX-1.1 | Subjects Excluded From Analysis Set (Randomized Subjects) |
| SUBEX-1.2 | Subjects Excluded From Analysis Set (Non-randomized Subjects) |